CLINICAL TRIAL: NCT00162266
Title: A Phase IIB, Multi-Center, Randomized, Double-Blind, Placebo Controlled Study to Evaluate the Safety and Clinical Efficacy of Two Different Doses of BMS-188667 Administered Intravenously to Subjects With Active Rheumatoid Arthritis While Receiving Methotrexate
Brief Title: Abatacept With Methotrexate- Phase IIB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM101-100
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Results first posted 2012-06-01 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Abatacept (10 mg/Kg) - Open Label (Experimental)
  Interventions: Drug: Abatacept (BMS-188667)
- Abatacept (2 mg/kg) - Double blind (Experimental)
  Interventions: Drug: Abatacept (BMS-188667)
- Abatacept (10 mg/kg) - Double blind (Experimental)
  Interventions: Drug: Abatacept (BMS-188667)
- Placebo - Double blind (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Abatacept (BMS-188667) — IV, 10 mg/Kg, monthly, for the duration of the trial
  Arms: Abatacept (10 mg/Kg) - Open Label
Drug: Abatacept (BMS-188667) — Intravenous (IV) infusion, 2 mg/kg, infused intravenously for approximately 30 min, infusions on Days 1, 15, 30 and monthly thereafter for 12 months
  Arms: Abatacept (2 mg/kg) - Double blind
Drug: Abatacept (BMS-188667) — Intravenous (IV) infusion, 10 mg/kg, infused intravenously for approximately 30 min, infusions on Days 1, 15, 30 and monthly thereafter for 12 months
  Arms: Abatacept (10 mg/kg) - Double blind
Drug: Placebo — Intravenous (IV) infusion, 0 mg/kg, infused intravenously for approximately 30 min, infusions on Days 1, 15, 30 and monthly thereafter for 12 months
  Arms: Placebo - Double blind

SUMMARY:
This study was conducted to assess the safety and tolerability of Abatacept combined with Methotrexate in participants with active rheumatoid arthritis (RA). The secondary objectives were to assess efficacy, pharmacodynamic marker activity, and immunogenicity of Abatacept combined with Methotrexate.

DETAILED DESCRIPTION:
All participants who completed the 12-month double-blind study period were eligible to continue in the open-label study. Participants received placebo, Abatacept 2 mg/kg, or Abatacept 10 mg/kg in the double-blind study. Participants receiving placebo in the double-blind study were switched 1:1 to continued treatment with placebo or Abatacept 2 mg/kg. Participants receiving Abatacept 2 mg/kg or Abatacept 10 mg/kg continued at the double-blind study dosage. After results from the double-blind period became available, all participants were switched to a weight-tiered 10 mg/kg dose of Abatacept.

Open label study design: Single group assignment, Single arm, Open label,

ELIGIBILITY:
Inclusion Criteria:

Double blind study phase:

1. Males or females (not nursing and not pregnant), at least 18 years of age. Women of child bearing potential (WOCBP) are eligible if they are practicing effective contraceptive measures
2. Subjects must meet the criteria of the American Rheumatism Association (1987) for the diagnosis of rheumatoid arthritis and the American College of Rheumatology (1991) functional classes I, II, or III
3. Subjects have been taking Methotrexate (10-30 mg weekly) for at least 6 months, and at a stable dose for 28 days prior to treatment
4. Washout/drug stabilization requirements (except Methotrexate) [Informed consent must be signed before making any changes in RA therapy if those changes are solely for the purpose of this study].

   * Leflunomide or Infliximab have already been discontinued at least 60 days prior to enrollment (prior to signing of informed consent) and a total of 90 days prior to treatment. All other Disease Modifying Anti-Rheumatic Drugs (DMARDs) (except Methotrexate) have been withdrawn at least 28 days prior to treatment
   * Oral corticosteroid treatment has been reduced to the equivalent of 10 mg or less prednisone daily and stabilized for at least 28 days prior to enrollment
5. Eligibility of subjects for the study is based on their disease activity and anti-rheumatic treatment at the initial visit:

   * Methotrexate monotherapy: Subject is receiving only Methotrexate, steroids, Non-steroidal anti-inflammatory drugs (NSAIDs) and will not require washout
   * Combination therapy: Subject is receiving Methotrexate in combination with another DMARD(s) and will require washout

   At entry, Methotrexate monotherapy must have a disease activity:
   * 10 or more swollen joints (66 joint count)
   * 12 or more tender joints (68 joint count)
   * C reactive protein (CRP) ≥.1 mg/dL (10 mg/L) at "Screening" visit

   At entry, combination therapy must have a disease activity (if subject does not satisfy the above):
   * 6 or more swollen joints (66 joint count)
   * 8 or more tender joints (68 joint count)
   * No restriction on C-reactive protein (CRP)

   In addition

   All subjects who were on combination therapy at entry must undergo a 28 day washout period of DMARDs other than Methotrexate. After the washout/drug stabilization and prior to randomization such subjects must have:
   * 10 or more swollen joints (66 joint count)
   * 12 or more tender joints (68 joint count)
   * C reactive protein (CRP) ≥ 1 mg/dL (10 mg/L)
6. Subject is willing to participate in the study and willing to sign the informed consent

Open label study phase:

* Participants that have completed the initial short term portion (double blind) of the study

Exclusion Criteria:

Double blind study phase:

1. Subjects who have at any time received treatment with BMS-188667 (Abatacept)
2. Subjects who within 30 days of the Day 1 visit have received treatment with any investigational drug
3. Subjects with active vasculitis of a major organ system (except for subcutaneous rheumatoid nodules)
4. Current symptoms of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, pulmonary, cardiac, neurological, or cerebral disease. Concomitant medical conditions that in the opinion of the investigator might place the subject at unacceptable risk for participation in this study
5. Mammogram requiring further investigation or biopsies leading to the diagnosis of a clinically significant abnormality. Complete evaluation of lesion is required before initiation of dosing
6. Subjects with a history of cancer within the last five years (other than non-melanoma skin cell cancers cured by local resection)
7. Subjects who have a history of clinically significant drug or alcohol abuse, or admit to consumption of more than 1 alcoholic drink per day
8. Subjects with evidence (as assessed by the investigator) of active or latent bacterial or viral infections at the time of potential enrollment, including subjects with evidence of Human Immunodeficiency Virus (HIV) infection, or hepatitis B or C infection
9. Subjects with any serious or chronic infections such as pneumonia, pyelo-nephritis, renal infection, chest infection with bronchiectasis, or sinusitis in the previous 3 months
10. Subjects with active tuberculosis requiring treatment within the previous 3 years
11. Subjects with any opportunistic infections such as herpes zoster or cytomegalovirus (CMV) within the previous 2 months
12. Subjects with severe asthma defined as > 3 emergency room admissions in the last year or > 3 treatments with oral steroids for asthma in the last year
13. A history of either angioedema or anaphylaxis that was associated with a reaction to a drug
14. Subjects with the following laboratory values:

    * Hemoglobin < 8.5 g/dL
    * White blood cells < 3000/mm3
    * Platelets < 100,000/mm3
    * Serum creatinine > 2 times upper limit of normal
    * Serum Alanine aminotransferase (ALAT) or Aspartate aminotransferase (ASAT) > 2 times upper limit of normal
    * Any other lab values that in the opinion of the investigator might place the subject at unacceptable risk for participation in this study

Open label study phase:

* Participants must continue to meet inclusion/exclusion criteria as in the short term (double blind) phase of the protocol except subjects who have receiving other than Abatacept

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Actual)
Dates: Start 2000-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (57):
- United States (26):
  - Local Institution, Birmingham, Alabama
  - Local Institution, Huntsville, Alabama
  - Local Institution, Long Beach, California
  - Local Institution, Highlands Ranch, Colorado
  - Local Institution, Largo, Florida
  - Local Institution, Titusville, Florida
  - Local Institution, West Palm Beach, Florida
  - Local Institution, Rome, Georgia
  - Local Institution, Chicago, Illinois
  - Local Institution, Wichita, Kansas
  - Local Institution, Cumberland, Maryland
  - Local Institution, Springfield, Massachusetts
  - Local Institution, Worcester, Massachusetts
  - Local Institution, Duluth, Minnesota
  - Local Institution, Lincoln, Nebraska
  - Local Institution, Albuquerque, New Mexico
  - Local Institution, Los Alamos, New Mexico
  - Local Institution, Albany, New York
  - Local Institution, Binghamton, New York
  - Local Institution, The Bronx, New York
  - Local Institution, Portland, Oregon
  - Local Institution, Duncansville, Pennsylvania
  - Local Institution, Sellersville, Pennsylvania
  - Local Institution, Amarillo, Texas
  - Local Institution, Austin, Texas
  - Local Institution, Dallas, Texas
- Argentina (2):
  - Local Institution, Buenos Aries, Buenos Aries
  - Local Institution, Quilmes, Burenos Aires
- Australia (3):
  - Local Institution, Adelaide, South Australia
  - Local Institution, Malvern, Victoria
  - Local Institution, Perth, Western Australia
- Belgium (5):
  - Local Institution, Antwerp
  - Local Institution, Brussels
  - Local Institution, Ghent
  - Local Institution, Leuven
  - Local Institution, Mons
- Canada (7):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Ottawa, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec
  - Local Institution, Sherbrooke, Quebec
  - Local Institution, Ste-Foy, Quebec
  - Local Institution, St. John's
- France (3):
  - Local Institution, Montpellier, Cedex
  - Local Institution, Strasbourg, Cedex
  - Local Institution, Paris
- Germany (3):
  - Local Institution, Berlin
  - Local Institution, Freiburg im Breisgau
  - Local Institution, Jena
- Local Institution, Cork, Cork, Ireland
- Local Institution, Nijmegen, Netherlands
- South Africa (2):
  - Local Institution, Muckleneuk, Gauteng
  - Local Institution, Cape Town, Western Cape
- United Kingdom (4):
  - Local Institution, Cambridge, Cambridgeshire
  - Local Institution, Manchester, Greater Manchester
  - Local Institution, Maidstone, Kent
  - Local Institution, Leeds, Yorkshire

REFERENCES:
- [Derived] Westhovens R, Kremer JM, Emery P, Russell AS, Alten R, Barre E, Dougados M. Long-term safety and efficacy of abatacept in patients with rheumatoid arthritis and an inadequate response to methotrexate: a 7-year extended study. Clin Exp Rheumatol. 2014 Jul-Aug;32(4):553-62. Epub 2014 Jul 8. PMID 25005467

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 524 subjects who were enrolled in this study, 185 were not randomized (1 reason unknown; 2 adverse event; 9 withdrawal of consent; 160 failure to meet inclusion and/or exclusion criteria; 1 death; 12 for other reasons).
Groups:
- Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX): Participants in the DB study received a weight-tiered dose of 10 mg/kg of abatacept that was administered monthly by an intravenous (IV) plus methotrexate (MTX).Participants were maintained on a stable dose of MTX (10-30 mg/wk) during Days 1 to 180 of the DB period; adjustments in corticosteroids (maximum 10 mg/day) and MTX (maximum 30 mg/wk) were permitted (as well as addition of either hydroxychloroquine, sulfasalazine, gold or azathioprine) during Days 181 to 360 of the DB period.
- Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate: Participants in the DB study received a weight-tiered dose of 2 mg/kg of abatacept that was administered monthly by an intravenous (IV) plus methotrexate (MTX).Participants were maintained on a stable dose of MTX (10-30 mg/wk) during Days 1 to 180 of the DB period; adjustments in corticosteroids (maximum 10 mg/day) and MTX (maximum 30 mg/wk) were permitted (as well as addition of either hydroxychloroquine, sulfasalazine, gold or azathioprine) during Days 181 to 360 of the DB period.
- Double-Blind (DB) Placebo + Methotrexate: Participants in the DB study received a placebo that was administered monthly by an intravenous (IV) plus methotrexate (MTX).Participants were maintained on a stable dose of MTX (10-30 mg/wk) during Days 1 to 180 of the DB period; adjustments in corticosteroids (maximum 10 mg/day) and MTX (maximum 30 mg/wk) were permitted (as well as addition of either hydroxychloroquine, sulfasalazine, gold or azathioprine) during Days 181 to 360 of the DB period.
- Open-Label (OL) Abatacept (10 mg / kg): Following a 5-month interim (where the placebo group was split into 2mg/kg abatacept or placebo and participants in 2 original abatacept continued at same dose), participants who enrolled in OL period received a weight-tiered dose of 10 mg/kg of abatacept that was administered monthly by an intravenous (IV) infusion over approximately 30 minutes. Participants weighing < 60 kg received abatacept 500 mg, participants weighing ≥ 60 kg and ≤ 100 kg received abatacept 750 mg, and participants > 100 kg received abatacept 1 g.
Period: Double-Blind Period
Arm/Group | Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) | Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate | Double-Blind (DB) Placebo + Methotrexate | Open-Label (OL) Abatacept (10 mg / kg)
Started | 115 | 105 | 119 | 0
Completed Day 1 to Day 181 | 98 | 80 | 78 | 0
Completed | 90 | 74 | 71 | 0
Not Completed | 25 | 31 | 48 | 0
Not completed — Adverse Event | 5 | 9 | 11 | 0
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0
Not completed — Other Reason | 1 | 0 | 1 | 0
Not completed — Lack of Efficacy | 13 | 17 | 30 | 0
Not completed — Withdrawal by Subject | 5 | 2 | 6 | 0
Period: Open-Label Period
Arm/Group | Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) | Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate | Double-Blind (DB) Placebo + Methotrexate | Open-Label (OL) Abatacept (10 mg / kg)
Started | 0 | 0 | 0 | 219
Completed | 0 | 0 | 0 | 82
Not Completed | 0 | 0 | 0 | 137
Not completed — Death | 0 | 0 | 0 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 46
Not completed — Lack of Efficacy | 0 | 0 | 0 | 26
Not completed — Lost to Follow-up | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 31
Not completed — Administrative Reason By Sponsor | 0 | 0 | 0 | 9
Not completed — Other Reasons | 0 | 0 | 0 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) | Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate | Double-Blind (DB) Placebo + Methotrexate | Total
Number analyzed (Participants) | 115 | 105 | 119 | 339
Age Continuous [Mean (Standard Deviation); unit: years] | 55.8 (12.5) | 54.4 (11.3) | 54.7 (12.0) | 55.0 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 66 | 79 | 231
  Male | 29 | 39 | 40 | 108
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 100 | 91 | 104 | 295
  Black | 6 | 0 | 3 | 9
  Other | 9 | 14 | 12 | 35
Weight [Mean (Standard Deviation); unit: Kg] | 77.8 (18.6) | 78.7 (21.4) | 79.9 (17.6) | 78.8 (19.2)
Rheumatoid Factor Status [Number; unit: Participants] — Status was not recorded for 4 participants.
  Participants
    Negative | 14 | 15 | 27 | 56
    Positive | 99 | 90 | 90 | 279
Number of Tender Joints [Mean (Standard Deviation); unit: Joints] | 30.8 (12.2) | 28.2 (12.0) | 29.2 (13.0) | 29.4 (12.4)
Number of Swollen Joints [Mean (Standard Deviation); unit: Joints] | 21.3 (8.4) | 20.2 (8.9) | 21.8 (8.8) | 21.1 (8.7)
C-Reactive Protein (CRP) Serum Level [Mean (Standard Deviation); unit: mg/dL] | 2.9 (2.8) | 3.2 (2.5) | 3.2 (3.2) | 3.1 (2.9)
Duration of Participant Rheumatoid Arthritis (RA) [Mean (Standard Deviation); unit: Years] | 9.7 (9.8) | 9.7 (8.1) | 8.9 (8.3) | 9.4 (8.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders to American College of Rheumatology 20% Improvement Criteria (ACR 20) at Day 180 of the Double-Blind (DB) Period
Description: ACR 20 response requires a participant to have a 20% reduction in the number of swollen and tender joints, and a reduction of 20% in three of the following five parameters: physician global assessment of disease, participant global assessment of disease, participant assessment of pain, C-reactive protein or erythrocyte sedimentation rate, and degree of disability in Health Assessment Questionnaire score. A participant achieved a sustained ACR 20 response if the participant had ACR 20 observed for at least 2 consecutive study visits.
Time Frame: Day 180
Population: Intent-to-treat population. Participants who discontinued the study due to lack of efficacy (ie, worsening rheumatoid arthritis) were considered ACR 20 nonresponders at all subsequent time points. For all subjects who discontinued for other reasons, their last ACR 20 response was carried forward.
Measure: Number; unit: Participants
Groups:
- DB Abatacept 10 mg/kg + Methotrexate: Participants received a weight-tiered dose of 10 mg/kg of abatacept, administered intravenously(IV) monthly plus methotrexate. Participants were maintained on a stable dose of methotrexate(10-30 mg/wk) during Days 1 to 180 of the DB period; adjustments in corticosteroids (maximum 10 mg/day) and methotrexate (maximum 30 mg/wk) were permitted (as well as addition of either hydroxychloroquine, sulfasalazine, gold or azathioprine) during Days 181 to 360 of the DB period.
- DB Abatacept 2 mg/kg + Methotrexate: Participants in the DB study received a weight-tiered dose of 2 mg/kg of abatacept administered IV monthly plus methotrexate. Participants were maintained on a stable dose of methotrexate (10-30 mg/wk) during Days 1 to 180 of the DB period; adjustments in corticosteroids (maximum 10 mg/day) and methotrexate (maximum 30 mg/wk) were permitted (as well as addition of either hydroxychloroquine, sulfasalazine, gold, or azathioprine) during Days 181 to 360 of the DB period.
- DB Placebo + Methotrexate: Participants in the DB study received a placebo that was administered IV monthly plus methotrexate. Participants were maintained on a stable dose of methotrexate (10-30 mg/wk) during Days 1 to 180 of the DB period; adjustments in corticosteroids (maximum 10 mg/day) and methotrexate(maximum 30 mg/wk) were permitted (as well as addition of either hydroxychloroquine, sulfasalazine, gold, or azathioprine) during Days 181 to 360 of the DB period.
Arm/Group | DB Abatacept 10 mg/kg + Methotrexate | DB Abatacept 2 mg/kg + Methotrexate | DB Placebo + Methotrexate
Number analyzed (Participants) | 115 | 105 | 119
Participants | 70 | 44 | 42
Statistical Analysis 1: Comparison: DB Abatacept 10 mg/kg + Methotrexate vs DB Placebo + Methotrexate; Test type: Superiority or Other; p < 0.001, Chi-squared; Point Estimate of Difference = 25.6, 95% CI 2-sided [12.8 to 38.4]
Statistical Analysis 2: Comparison: DB Abatacept 2 mg/kg + Methotrexate vs DB Placebo + Methotrexate; Test type: Superiority or Other; p = 0.31, Chi-squared; Point Estimate of Difference = 6.6, 95% CI 2-sided [-6.2 to 19.4]

2. Secondary Outcome: Number of ACR 20 Responders in DB Period
Description: ACR 20 response requires a participant to have a 20% reduction in the number of swollen and tender joints, and a reduction of 20% in three of the following five parameters: physician global assessment of disease, participant global assessment of disease, participant assessment of pain, C-reactive protein or erythrocyte sedimentation rate, and degree of disability in HAQ score. A participant achieved a sustained ACR 20 response if the participant had ACR 20 observed for at least 2 consecutive study visits.
Time Frame: Days 15, 30, 60, 90, 120, 150,180, 240, 300, and 360
Population: Participants who received at least 1 infusion of study medication
Measure: Number; unit: Participants
Groups:
- DB Abatacept 10 mg/kg + Methotrexate: Participants in the DB study received a weight-tiered dose of 10 mg/kg of abatacept administered monthly IV plus methotrexateParticipants were maintained on a stable dose of methotrexate (10-30 mg/wk) during Days 1 to 180 of the DB period; adjustments in corticosteroids (maximum 10 mg/day) and methotrexate (maximum 30 mg/wk) were permitted (as well as addition of either hydroxychloroquine, sulfasalazine, gold or azathioprine) during Days 181 to 360 of the DB period.
- DB Abatacept 2 mg/kg + Methotrexate: Participants in the DB study received a weight-tiered dose of 2 mg/kg of abatacept administered monthly IV plus methotrexate. Participants were maintained on a stable dose of methotrexate(10-30 mg/wk) during Days 1 to 180 of the DB period; adjustments in corticosteroids (maximum 10 mg/day) and methotrexate (maximum 30 mg/wk) were permitted (as well as addition of either hydroxychloroquine, sulfasalazine, gold or azathioprine) during Days 181 to 360 of the DB period.
- DB Placebo + Methotrexate: Participants in the DB study received a placebo administered monthly IV plus methotrexate. Participants were maintained on a stable dose of methotrexate (10-30 mg/wk) during Days 1 to 180 of the DB period; adjustments in corticosteroids (maximum 10 mg/day) and methotrexate(maximum 30 mg/wk) were permitted (as well as addition of either hydroxychloroquine, sulfasalazine, gold or azathioprine) during Days 181 to 360 of the DB period.
Arm/Group | DB Abatacept 10 mg/kg + Methotrexate | DB Abatacept 2 mg/kg + Methotrexate | DB Placebo + Methotrexate
Number analyzed (Participants) | 115 | 105 | 119
Participants
  Day 15 | 30 | 9 | 24
  Day 30 | 48 | 22 | 36
  Day 60 | 65 | 35 | 41
  Day 90 | 62 | 40 | 42
  Day 120 | 71 | 47 | 45
  Day 150 | 67 | 46 | 42
  Day 180 | 70 | 44 | 42
  Day 240 | 72 | 43 | 42
  Day 300 | 73 | 41 | 41
  Day 360 | 72 | 44 | 43
Statistical Analysis 1: Comparison: DB Abatacept 10 mg/kg + Methotrexate vs DB Placebo + Methotrexate; Response on Day 15; Test type: Superiority or Other; p = 0.283, Chi-squared; Point Estimate of Difference = 5.9, 95% CI 2-sided [-4.9 to 16.7]
Statistical Analysis 2: Comparison: DB Abatacept 2 mg/kg + Methotrexate vs DB Placebo + Methotrexate; Response on Day 15; Test type: Superiority or Other; p = 0.015, Chi-squared; Point Estimate of Difference = -11.6, 95% CI 2-sided [-20.9 to -2.3]
Statistical Analysis 3: Comparison: DB Abatacept 10 mg/kg + Methotrexate vs DB Placebo + Methotrexate; Response on Day 30; Test type: Superiority or Other; p = 0.067, Chi-squared; Point Estimate of Difference = 11.5, 95% CI 2-sided [-0.8 to 23.8]
Statistical Analysis 4: Comparison: DB Abatacept 2 mg/kg + Methotrexate vs DB Placebo + Methotrexate; Response on Day 30; Test type: Superiority or Other; p = 0.113, Chi-squared; Point Estimate of Difference = -9.3, 95% CI 2-sided [-20.8 to 2.2]
Statistical Analysis 5: Comparison: DB Abatacept 10 mg/kg + Methotrexate vs DB Placebo + Methotrexate; Response on Day 60; Test type: Superiority or Other; p < 0.001, Chi-squared; Point Estimate of Difference = 22.1, 95% CI 2-sided [9.3 to 34.8]
Statistical Analysis 6: Comparison: DB Abatacept 2 mg/kg + Methotrexate vs DB Placebo + Methotrexate; Response on Day 60; Test type: Superiority or Other; p = 0.86, Chi-squared; Point Estimate of Difference = -1.1, 95% CI 2-sided [-13.5 to 11.3]
Statistical Analysis 7: Comparison: DB Abatacept 10 mg/kg + Methotrexate vs DB Placebo + Methotrexate; Response on Day 90; Test type: Superiority or Other; p = 0.004, Chi-squared; Point Estimate of Difference = 18.6, 95% CI 2-sided [5.9 to 31.4]
Statistical Analysis 8: Comparison: DB Abatacept 2 mg/kg + Methotrexate vs DB Placebo + Methotrexate; Response on Day 90; Test type: Superiority or Other; p = 0.664, Chi-squared; Point Estimate of Difference = 2.8, 95% CI 2-sided [-9.8 to 15.4]
Statistical Analysis 9: Comparison: DB Abatacept 10 mg/kg + Methotrexate vs DB Placebo + Methotrexate; Response on Day 120; Test type: Superiority or Other; p < 0.001, Chi-squared; Point Estimate of Difference = 23.9, 95% CI 2-sided [11.1 to 36.7]
Statistical Analysis 10: Comparison: DB Abatacept 2 mg/kg + Methotrexate vs DB Placebo + Methotrexate; Response on Day 120; Test type: Superiority or Other; p = 0.292, Chi-squared; Point Estimate of Difference = 6.9, 95% CI 2-sided [-6.0 to 19.9]
Statistical Analysis 11: Comparison: DB Abatacept 10 mg/kg + Methotrexate vs DB Placebo + Methotrexate; Response on Day 150; Test type: Superiority or Other; p < 0.001, Chi-squared; Point Estimate of Difference = 23.0, 95% CI 2-sided [10.2 to 35.8]
Statistical Analysis 12: Comparison: DB Abatacept 2 mg/kg + Methotrexate vs DB Placebo + Methotrexate; Response on Day 150; Test type: Superiority or Other; p = 0.193, Chi-squared; Point Estimate of Difference = 8.5, 95% CI 2-sided [-4.3 to 21.3]
Statistical Analysis 13: Comparison: DB Abatacept 10 mg/kg + Methotrexate vs DB Placebo + Methotrexate; Response on Day 180; Test type: Superiority or Other; p < 0.001, Chi-squared; Point Estimate of Difference = 25.6, 95% CI 2-sided [12.8 to 38.4]
Statistical Analysis 14: Comparison: DB Abatacept 2 mg/kg + Methotrexate vs DB Placebo + Methotrexate; Response on Day 180; Test type: Superiority or Other; p = 0.31, Chi-squared; Point Estimate of Difference = 6.6, 95% CI [-6.2 to 19.4]
Statistical Analysis 15: Comparison: DB Abatacept 10 mg/kg + Methotrexate vs DB Placebo + Methotrexate; Response on Day 240; Test type: Superiority or Other; p < 0.001, Chi-squared; Point Estimate of Difference = 27.3, 95% CI 2-sided [14.5 to 40.1]
Statistical Analysis 16: Comparison: DB Abatacept 2 mg/kg + Methotrexate vs DB Placebo + Methotrexate; Response on Day 240; Test type: Superiority or Other; p = 0.384, Chi-squared; Point Estimate of Difference = 5.7, 95% CI 2-sided [-7.1 to 18.4]
Statistical Analysis 17: Comparison: DB Abatacept 10 mg/kg + Methotrexate vs DB Placebo + Methotrexate; Response on Day 300; Test type: Superiority or Other; p < 0.001, Chi-squared; Point Estimate of Difference = 29.0, 95% CI 2-sided [16.2 to 41.8]
Statistical Analysis 18: Comparison: DB Abatacept 2 mg/kg + Methotrexate vs DB Placebo + Methotrexate; Response on Day 300; Test type: Superiority or Other; p = 0.476, Chi-squared; Point Estimate of Difference = 4.6, 95% CI 2-sided [-8.0 to 17.2]
Statistical Analysis 19: Comparison: DB Abatacept 10 mg/kg + Methotrexate vs DB Placebo + Methotrexate; Response on Day 360; Test type: Superiority or Other; p < 0.001, Chi-squared; Point Estimate of Difference = 26.5, 95% CI 2-sided [13.7 to 39.3]
Statistical Analysis 20: Comparison: DB Abatacept 2 mg/kg + Methotrexate vs DB Placebo + Methotrexate; Response on Day 360; Test type: Superiority or Other; p = 0.377, Chi-squared; Point Estimate of Difference = 5.8, 95% CI 2-sided [-7.0 to 18.6]

3. Secondary Outcome: Number of ACR 50 Responders in DB Period
Description: ACR 50 response requires a participant to have a 50% reduction in the number of swollen and tender joints, and a reduction of 50% in three of the following five parameters: physician global assessment of disease, participant global assessment of disease, participant assessment of pain, C-reactive protein or erythrocyte sedimentation rate, and degree of disability in HAQ score. A participant achieved a sustained ACR 50 response if the participant had ACR 50 observed for at least 2 consecutive study visits.
Time Frame: Day 15; Day 30; Day 60; Day 90; Day 120; Day 150; Day 180; Day 240; Day 300; Day 360
Population: Participants who received at least 1 infusion of study medication
Measure: Number; unit: Participants
Arm/Group | Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) | Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate | Double-Blind (DB) Placebo + Methotrexate
Number analyzed (Participants) | 115 | 105 | 119
Participants
  Day 15 | 2 | 0 | 3
  Day 30 | 16 | 4 | 7
  Day 60 | 25 | 14 | 18
  Day 90 | 28 | 18 | 15
  Day 120 | 38 | 18 | 18
  Day 150 | 42 | 18 | 19
  Day 180 | 42 | 24 | 14
  Day 240 | 41 | 22 | 24
  Day 300 | 45 | 23 | 18
  Day 360 | 48 | 24 | 24
Statistical Analysis 1: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 15; Test type: Superiority or Other; p = 0.679, Chi-squared; Point Estimate of Difference = -0.8, 95% CI 2-sided [-4.5 to 2.9]
Statistical Analysis 2: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 15; Test type: Superiority or Other; p = 0.101, Chi-squared; Point Estimate of Difference = -2.5, 95% CI 2-sided [-5.5 to 0.5]
Statistical Analysis 3: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 30; Test type: Superiority or Other; p = 0.039, Chi-squared; Point Estimate of Difference = 8.0, 95% CI 2-sided [0.4 to 15.7]
Statistical Analysis 4: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 30; Test type: Superiority or Other; p = 0.474, Chi-squared; Point Estimate of Difference = -2.1, 95% CI 2-sided [-7.7 to 3.6]
Statistical Analysis 5: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 60; Test type: Superiority or Other; p = 0.192, Chi-squared; Point Estimate of Difference = 6.6, 95% CI 2-sided [-3.3 to 16.5]
Statistical Analysis 6: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 60; Test type: Superiority or Other; p = 0.702, Chi-squared; Point Estimate of Difference = -1.8, 95% CI 2-sided [-11.0 to 7.4]
Statistical Analysis 7: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 90; Test type: Superiority or Other; p = 0.02, Chi-squared; Point Estimate of Difference = 11.7, 95% CI 2-sided [1.8 to 21.7]
Statistical Analysis 8: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 90; Test type: Superiority or Other; p = 0.339, Chi-squared; Point Estimate of Difference = 4.5, 95% CI 2-sided [-4.8 to 13.8]
Statistical Analysis 9: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 120; Test type: Superiority or Other; p = 0.001, Chi-squared; Point Estimate of Difference = 17.9, 95% CI 2-sided [7.0 to 28.9]
Statistical Analysis 10: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 120; Test type: Superiority or Other; p = 0.682, Chi-squared; Point Estimate of Difference = 2.0, 95% CI 2-sided [-7.6 to 11.7]
Statistical Analysis 11: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 150; Test type: Superiority or Other; p < 0.001, Chi-squared; Point Estimate of Difference = 20.6, 95% CI 2-sided [9.3 to 31.8]
Statistical Analysis 12: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 150; Test type: Superiority or Other; p = 0.813, Chi-squared; Point Estimate of Difference = 1.2, 95% CI 2-sided [-8.6 to 10.9]
Statistical Analysis 13: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 180; Test type: Superiority or Other; p < 0.001, Chi-squared; Point Estimate of Difference = 24.8, 95% CI 2-sided [13.8 to 35.7]
Statistical Analysis 14: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 180; Test type: Superiority or Other; p = 0.027, Chi-squared; Point Estimate of Difference = 11.1, 95% CI 2-sided [1.2 to 20.9]
Statistical Analysis 15: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 240; Test type: Superiority or Other; p = 0.008, Chi-squared; Point Estimate of Difference = 15.5, 95% CI 2-sided [4.0 to 27.0]
Statistical Analysis 16: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 240; Test type: Superiority or Other; p = 0.885, Chi-squared; Point Estimate of Difference = 0.8, 95% CI 2-sided [-9.8 to 11.4]
Statistical Analysis 17: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 300; Test type: Superiority or Other; p < 0.001, Chi-squared; Point Estimate of Difference = 24.0, 95% CI 2-sided [12.6 to 35.4]
Statistical Analysis 18: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 300; Test type: Superiority or Other; p = 0.19, Chi-squared; Point Estimate of Difference = 6.8, 95% CI 2-sided [-3.4 to 16.9]
Statistical Analysis 19: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 360; Test type: Superiority or Other; p < 0.001, Chi-squared; Point Estimate of Difference = 21.6, 95% CI 2-sided [9.7 to 33.4]
Statistical Analysis 20: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 360; Test type: Superiority or Other; p = 0.625, Chi-squared; Point Estimate of Difference = 2.7, 95% CI 2-sided [-8.1 to 13.5]

4. Secondary Outcome: Number of ACR 70 Responders in DB Period
Description: ACR 70 response requires a participant to have a 70% reduction in the number of swollen and tender joints, and a reduction of 70% in three of the following five parameters: physician global assessment of disease, participant global assessment of disease, participant assessment of pain, C-reactive protein or erythrocyte sedimentation rate, and degree of disability in HAQ score. A participant achieved a sustained ACR 70 response if the participant had ACR 70 observed for at least 2 consecutive study visits.
Time Frame: Day 15; Day 30; Day 60; Day 90; Day 120; Day 150; Day 180; Day 240; Day 300; Day 360
Population: Participants who received at least 1 infusion of study medication
Measure: Number; unit: Participants
Arm/Group | Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) | Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate | Double-Blind (DB) Placebo + Methotrexate
Number analyzed (Participants) | 115 | 105 | 119
Participants
  Day 15 | 0 | 0 | 0
  Day 30 | 4 | 3 | 0
  Day 60 | 10 | 4 | 0
  Day 90 | 10 | 5 | 1
  Day 120 | 15 | 6 | 4
  Day 150 | 16 | 6 | 4
  Day 180 | 19 | 11 | 2
  Day 240 | 21 | 9 | 6
  Day 300 | 27 | 11 | 3
  Day 360 | 24 | 13 | 9
Statistical Analysis 1: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 30; Test type: Superiority or Other; p = 0.04, Chi-squared; Point Estimate of Difference = 3.5, 95% CI [0.2 to 6.8]
Statistical Analysis 2: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 30; Test type: Superiority or Other; p = 0.063, Chi-squared; Point Estimate of Difference = 2.9, 95% CI 2-sided [-0.2 to 5.9]
Statistical Analysis 3: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 60; Test type: Superiority or Other; p = 0.001, Chi-squared; Point Estimate of Difference = 8.7, 95% CI 2-sided [3.5 to 13.9]
Statistical Analysis 4: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 60; Test type: Superiority or Other; p = 0.032, Chi-squared; Point Estimate of Difference = 3.8, 95% CI 2-sided [0.3 to 7.3]
Statistical Analysis 5: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 90; Test type: Superiority or Other; p = 0.005, Chi-squared; Point Estimate of Difference = 7.9, 95% CI 2-sided [2.4 to 13.3]
Statistical Analysis 6: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 90; Test type: Superiority or Other; p = 0.07, Chi-squared; Point Estimate of Difference = 3.9, 95% CI 2-sided [-0.3 to 8.2]
Statistical Analysis 7: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 120; Test type: Superiority or Other; p = 0.007, Chi-squared; Point Estimate of Difference = 9.7, 95% CI 2-sided [2.7 to 16.7]
Statistical Analysis 8: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Test type: Superiority or Other; p = 0.395, Chi-squared; Point Estimate of Difference = 2.4, 95% CI [-3.1 to 7.8]
Statistical Analysis 9: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 150; Test type: Superiority or Other; p = 0.004, Chi-squared; Point Estimate of Difference = 10.6, 95% CI 2-sided [3.4 to 17.7]
Statistical Analysis 10: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 150; Test type: Superiority or Other; p = 0.395, Chi-squared; Point Estimate of Difference = 2.4, 95% CI 2-sided [-3.1 to 7.8]
Statistical Analysis 11: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 180; Test type: Superiority or Other; p < 0.001, Chi-squared; Point Estimate of Difference = 14.8, 95% CI 2-sided [7.5 to 22.2]
Statistical Analysis 12: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 180; Test type: Superiority or Other; p = 0.005, Chi-squared; Point Estimate of Difference = 8.8, 95% CI 2-sided [2.7 to 14.9]
Statistical Analysis 13: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 240; Test type: Superiority or Other; p = 0.002, Chi-squared; Point Estimate of Difference = 13.2, 95% CI 2-sided [5.0 to 21.4]
Statistical Analysis 14: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 240; Test type: Superiority or Other; p = 0.292, Chi-squared; Point Estimate of Difference = 3.5, 95% CI 2-sided [-3.0 to 10.1]
Statistical Analysis 15: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 300; Test type: Superiority or Other; p < 0.001, Chi-squared; Point Estimate of Difference = 21.0, 95% CI 2-sided [12.4 to 29.5]
Statistical Analysis 16: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 300; Test type: Superiority or Other; p = 0.014, Chi-squared; Point Estimate of Difference = 8.0, 95% CI 2-sided [1.6 to 14.3]
Statistical Analysis 17: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 360; Test type: Superiority or Other; p = 0.003, Chi-squared; Point Estimate of Difference = 13.3, 95% CI 2-sided [4.4 to 22.2]
Statistical Analysis 18: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Response on Day 360; Test type: Superiority or Other; p = 0.227, Chi-squared; Point Estimate of Difference = 4.8, 95% CI 2-sided [-3.0 to 12.6]

5. Secondary Outcome: ACR Numeric Values (ACR-N)
Description: The ACR-N is calculated for each participant by taking the lowest percentage improvement in (1) swollen joint count or (2) tender joint count or (3) the median of the remaining 5 components of the ACR response (participant's assessment of disease activity; participant's global assessment of pain; physician's assessment of disease activity; participant's assessment of physical function; an acute phase reactant value - CRP). Negative numbers indicate worsening.
Time Frame: Day 15; Day 30; Day 60; Day 90; Day 120; Day 150; Day 180; Day 240; Day 300; Day 360
Population: Participants who received at least 1 infusion of study medication
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) | Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate | Double-Blind (DB) Placebo + Methotrexate
Number analyzed (Participants) | 115 | 105 | 119
units on a scale
  Day 15 (n=113, 104, 118) | 11.09 (15.53) | 5.26 (10.37) | 9.07 (14.76)
  Day 30 (n=115, 104, 117) | 20.45 (23.41) | 12.06 (18.11) | 13.20 (17.85)
  Day 60 (n=114, 105, 119) | 28.85 (26.78) | 17.69 (22.83) | 17.09 (20.90)
  Day 90 (n=115, 105, 118) | 29.03 (27.38) | 21.12 (26.10) | 16.93 (21.61)
  Day 120 (n=114, 105, 115) | 33.80 (29.35) | 22.87 (26.10) | 19.26 (23.70)
  Day 150 (n=114, 103, 118) | 36.34 (30.29) | 22.69 (24.15) | 19.37 (24.74)
  Day 180 (n=114, 104, 118) | 37.65 (30.39) | 24.67 (29.03) | 17.29 (22.02)
  Day 240 (n=115, 104, 119) | 38.34 (31.49) | 23.49 (27.51) | 20.71 (25.97)
  Day 300 (n=114, 105, 119) | 39.69 (31.08) | 21.82 (27.99) | 18.69 (23.53)
  Day 360 (n=115, 105, 119) | 40.87 (31.69) | 24.55 (29.37) | 20.49 (26.14)
Statistical Analysis 1: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Day 15 Treatment Comparison; Test type: Superiority or Other; p = 0.2676, ANOVA; ANOVA model: AUC = treatment; Mean Difference (Final Values) = 2.02, 95% CI 2-sided [-1.56 to 5.61] — Estimate= Model AUC for abatacept+methotrexate - Model AUC for placebo+methotrexate
Statistical Analysis 2: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Day 15 Treatment Comparison; Test type: Superiority or Other; p = 0.0418, ANOVA; ANOVA model: AUC = treatment; Mean Difference (Final Values) = -3.80, 95% CI 2-sided [-7.46 to -0.14] — Estimate= Model AUC for abatacept+methotrexate - Model AUC for placebo+methotrexate
Statistical Analysis 3: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Day 30 Treatment Comparison; Test type: Superiority or Other; p = 0.0061, ANOVA; ANOVA model: AUC = treatment; Mean Difference (Final Values) = 7.25, 95% CI 2-sided [2.08 to 12.41] — Estimate= Model AUC for abatacept+methotrexate - Model AUC for placebo+methotrexate
Statistical Analysis 4: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Day 30 Treatment Comparison; Test type: Superiority or Other; p = 0.6713, ANOVA — ANOVA model: AUC = treatment; Mean Difference (Final Values) = -1.14, 95% CI 2-sided [-6.45 to 4.16] — Estimate= Model AUC for abatacept+methotrexate - Model AUC for placebo+methotrexate
Statistical Analysis 5: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Day 60 Treatment Comparison; Test type: Superiority or Other; p = 0.0002, ANOVA; ANOVA model: AUC = treatment; Mean Difference (Final Values) = 11.75, 95% CI 2-sided [5.67 to 17.84] — Estimate= Model AUC for abatacept+methotrexate - Model AUC for placebo+methotrexate
Statistical Analysis 6: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Day 60 Treatment Comparison; Test type: Superiority or Other; p = 0.8495, ANOVA; ANOVA model: AUC = treatment; Mean Difference (Final Values) = 0.60, 95% CI 2-sided [-5.62 to 6.82] — Estimate= Model AUC for abatacept+methotrexate - Model AUC for placebo+methotrexate
Statistical Analysis 7: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Day 90 Treatment Comparison; Test type: Superiority or Other; p = 0.0003, ANOVA; ANOVA model: AUC = treatment; Mean Difference (Final Values) = 12.10, 95% CI 2-sided [5.63 to 18.56] — Estimate= Model AUC for abatacept+methotrexate - Model AUC for placebo+methotrexate
Statistical Analysis 8: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Day 90 Treatment Comparison; Test type: Superiority or Other; p = 0.0003, ANOVA; ANOVA model: AUC = treatment; Mean Difference (Final Values) = 4.19, 95% CI 2-sided [-2.44 to 10.81] — Estimate= Model AUC for abatacept+methotrexate - Model AUC for placebo+methotrexate
Statistical Analysis 9: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Day 120 Treatment Comparison; Test type: Superiority or Other; p = 0.0001, ANOVA; ANOVA model: AUC = treatment; Mean Difference (Final Values) = 14.54, 95% CI 2-sided [7.28 to 21.81] — Estimate= Model AUC for abatacept+methotrexate - Model AUC for placebo+methotrexate
Statistical Analysis 10: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Day 120 Treatment Comparison; Test type: Superiority or Other; p = 0.3141, ANOVA; ANOVA model: AUC = treatment; Mean Difference (Final Values) = 3.60, 95% CI 2-sided [-3.43 to 10.64] — Estimate= Model AUC for abatacept+methotrexate - Model AUC for placebo+methotrexate
Statistical Analysis 11: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Day 150 Treatment Comparison; Test type: Superiority or Other; p = 0.0001, ANOVA; ANOVA model: AUC = treatment; Mean Difference (Final Values) = 16.96, 95% CI 2-sided [8.49 to 25.43] — Estimate= Model AUC for abatacept+methotrexate - Model AUC for placebo+methotrexate
Statistical Analysis 12: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Day 150 Treatment Comparison; Test type: Superiority or Other; p = 0.3552, ANOVA; ANOVA model: AUC = treatment; Mean Difference (Final Values) = 3.32, 95% CI 2-sided [-3.73 to 10.37] — Estimate= Model AUC for abatacept+methotrexate - Model AUC for placebo+methotrexate
Statistical Analysis 13: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Day 180 Treatment Comparison; Test type: Superiority or Other; p = 0.0001, ANOVA; ANOVA model: AUC = treatment; Mean Difference (Final Values) = 20.36, 95% CI 2-sided [10.19 to 30.54] — Estimate= Model AUC for abatacept+methotrexate - Model AUC for placebo+methotrexate
Statistical Analysis 14: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Day 180 Treatment Comparison; Test type: Superiority or Other; p = 0.0451, ANOVA; ANOVA model: AUC = treatment; Mean Difference (Final Values) = 7.38, 95% CI 2-sided [0.16 to 14.60] — Estimate= Model AUC for abatacept+methotrexate - Model AUC for placebo+methotrexate
Statistical Analysis 15: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Day 240 Treatment Comparison; Test type: Superiority or Other; p = 0.0001, ANOVA; ANOVA model: AUC = treatment; Mean Difference (Final Values) = 17.63, 95% CI 2-sided [8.83 to 26.44] — Estimate= Model AUC for abatacept+methotrexate - Model AUC for placebo+methotrexate
Statistical Analysis 16: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Day 240 Treatment Comparison; Test type: Superiority or Other; p = 0.4669, ANOVA; ANOVA model: AUC = treatment; Mean Difference (Final Values) = 2.78, 95% CI 2-sided [-4.73 to 10.28] — Estimate= Model AUC for abatacept+methotrexate - Model AUC for placebo+methotrexate
Statistical Analysis 17: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Day 300 Treatment Comparison; Test type: Superiority or Other; p = 0.0001, ANOVA; ANOVA model: AUC = treatment; Mean Difference (Final Values) = 21.00, 95% CI 2-sided [10.51 to 31.48] — Estimate= Model AUC for abatacept+methotrexate - Model AUC for placebo+methotrexate
Statistical Analysis 18: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Day 300 Treatment Comparison; Test type: Superiority or Other; p = 3.13, ANOVA; ANOVA model: AUC = treatment; Mean Difference (Final Values) = 3.13, 95% CI 2-sided [-4.15 to 10.41] — Estimate= Model AUC for abatacept+methotrexate - Model AUC for placebo+methotrexate
Statistical Analysis 19: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Day 360 Treatment Comparison; Test type: Superiority or Other; p = 0.0001, ANOVA; ANOVA model: AUC = treatment; Mean Difference (Final Values) = 20.38, 95% CI 2-sided [10.20 to 30.56] — Estimate= Model AUC for abatacept+methotrexate - Model AUC for placebo+methotrexate
Statistical Analysis 20: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Day 360 Treatment Comparison; Test type: Superiority or Other; p = 0.2989, ANOVA; ANOVA model: AUC = treatment; Mean Difference (Final Values) = 4.06, 95% CI 2-sided [-3.61 to 11.72] — Estimate= Model AUC for abatacept+methotrexate - Model AUC for placebo+methotrexate

6. Secondary Outcome: ACR-N Area Under The Curve (AUC) on Day 180 and Day 360
Description: The AUC for ACR-N is the measure of the area under the curve of the mean change from baseline in ACR-N. The trapezoidal rule was used to compute the AUC. The ACR-N AUC was compared between the two abatacept treatment groups and the placebo group using an analysis of variance (ANOVA) for 6- and 12-month data (Day 180 and Day 360). This allowed for the assessment of subject response throughout the study. See Measure Description in Outcome Measure 18 for a definition of ACR-N.
Time Frame: Baseline and Day 180; Baseline and Day 360
Measure: Mean (Standard Error); unit: percentage*days
Arm/Group | Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) | Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate | Double-Blind (DB) Placebo + Methotrexate
Number analyzed (Participants) | 115 | 105 | 119
percentage*days
  Day 180 | 5021.70 (317.9) | 3242.54 (332.7) | 2889.07 (312.5)
  Day 360 | 12035.1 (711.7) | 7447.87 (744.8) | 6393.49 (699.6)
Statistical Analysis 1: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Comparison at Day 180; Test type: Superiority or Other; p = 0.0001, ANOVA — ANOVA model: AUC = treatment; Mean Difference (Final Values) = 2132.63, 95% CI 2-sided [1067.32 to 3197.94] — Estimate = Model AUC for Aripiprazole+MTX - Model AUC for PLACEBO+MTX
Statistical Analysis 2: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Comparison at Day 180; Test type: Superiority or Other; p = 0.4393, ANOVA — ANOVA model: AUC = treatment; Mean Difference (Final Values) = 353.47, 95% CI 2-sided [-544.46 to 1251.41] — Estimate = Model AUC for Aripiprazole+MTX - Model AUC for PLACEBO+MTX
Statistical Analysis 3: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Comparison at Day 360; Test type: Superiority or Other; p = 0.0001, ANOVA — ANOVA model: AUC = treatment; Mean Difference (Final Values) = 5641.60, 95% CI 2-sided [2823.46 to 8459.74] — Estimate = Model AUC for Aripiprazole+MTX - Model AUC for PLACEBO+MTX
Statistical Analysis 4: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Comparison at Day 360; Test type: Superiority or Other; p = 0.3029, ANOVA — ANOVA model: AUC = treatment; Mean Difference (Final Values) = 1054.38, 95% CI 2-sided [-955.59 to 3064.35] — Estimate = Model AUC for Aripiprazole+MTX - Model AUC for PLACEBO+MTX

7. Secondary Outcome: Individual Components of ACR Criteria--Mean Percentage Change From Baseline at Day 180
Description: Percentage change = 100*(Baseline value - value at specific visit) / Baseline value. The American College of Rheumatology (ACR) response criteria, based on a core set of variables which includes a tender joint count, a swollen joint count, patient-reported pain scale (Subject Assessment of Physical Function [SAPF]), patient and physician global assessments of disease activity (Subject Global Assessment [SGA] and Physician Global Assessment [PGA]), patient assessment of functional ability, and an acute phase reactant (C-Reactive Protein [CRP])
Time Frame: Baseline, Day 180
Population: Number of Participants Analyzed = Participants who received at least 1 infusion of study medication; n = subset of participants who had given measurement at both time points.
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) | Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate | Double-Blind (DB) Placebo + Methotrexate
Number analyzed (Participants) | 115 | 105 | 119
percentage change
  Tender Joints (n=114, 104, 118) | 59.8 (3.6) | 43.2 (4.1) | 31.9 (5.0)
  Swollen Joints (n=114, 104, 118) | 55.3 (3.5) | 45.3 (4.1) | 33.5 (4.3)
  Pain (n=109, 102, 118) | 46.2 (4.1) | 22.1 (5.8) | 8.2 (7.0)
  SAPF (n=107, 98, 110) | 41.2 (4.6) | 21.6 (6.5) | 13.7 (5.5)
  Subject Global Assessment (n=111, 103, 118) | 40.8 (4.7) | 9.1 (10.4) | 17.5 (4.1)
  Physician Global Assessment (n=111, 103, 116) | 51.9 (3.4) | 38.7 (4.4) | 25.1 (3.5)
  C-Reactive Protein (n=108, 98, 114) | 31.8 (6.3) | 16.4 (7.0) | -23.4 (11.0)

8. Secondary Outcome: Individual Components of ACR Criteria--Mean Percentage Change From Baseline at Day 360
Description: as for outcome 7
Time Frame: Baseline, Day 360
Population: as for outcome 7
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) | Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate | Double-Blind (DB) Placebo + Methotrexate
Number analyzed (Participants) | 115 | 105 | 119
percentage change
  Tender Joints (n=114, 104, 118) | 66.4 (3.8) | 43.6 (4.3) | 30.0 (5.3)
  Swollen Joints (n=114, 104, 118) | 59.7 (3.7) | 46.4 (4.5) | 36.2 (4.4)
  Pain (n=109, 102, 118) | 44.9 (4.7) | 26.2 (5.9) | 65.2 (12.6)
  SAPF (n=107, 98, 110) | 42.3 (4.3) | 22.9 (5.0) | 10.3 (5.9)
  Subject Global Assessment (n=111, 103, 118) | 41.0 (5.1) | 16.0 (8.9) | 2.0 (19.1)
  Physician Global Assessment (n=111, 103, 116) | 53.5 (3.4) | 37.9 (4.2) | 24.1 (3.8)
  C-Reactive Protein (n=108, 98, 114) | 27.6 (9.9) | 11.0 (9.5) | -31.3 (12.6)

9. Secondary Outcome: Mean Changes From Baseline in the Short Form 36 (SF-36) Physical and Mental Health Component Summary Scores (PCS and MCS) at Day 180 and Day 360
Description: SF-36 measures health-related quality of life across multiple disease states. It has 36 questions with 8 subscale scores and 2 summary scores: PCS=physical functioning, role-physical, bodily pain, and general health; MCS=vitality, social functioning, role-emotional, and mental health. Scoring is done for both subscores and summary scores. For both, 0=worst score (or quality of life) and 100=best score.
Time Frame: Baseline, Day 180, Day 360
Population: Number of Participants Analyzed=total number of participants in each treatment group. n=number of treated Participants with measurement at baseline and given timepoint.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) | Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate | Double-Blind (DB) Placebo + Methotrexate
Number analyzed (Participants) | 115 | 105 | 119
units on a scale
  PCS, Mean Change at Day 180 (n=115, 104, 119) | 8.3 (0.9) | 4.6 (0.7) | 3.0 (0.6)
  MCS, Mean Change at Day 180 (n=115, 104, 119) | 5.0 (1.0) | 2.7 (1.2) | 3.2 (1.0)
  PCS, Mean Change at Day 360 (n=115, 104, 119) | 8.1 (0.9) | 5.3 (0.8) | 2.8 (0.7)
  PCS, Mean Change at Day 360 (n=115, 104, 119) | 5.7 (1.0) | 3.5 (1.1) | 3.0 (0.9)

10. Secondary Outcome: Adjusted Mean Percent Changes From Baseline in the Modified Health Assessment Questionnaire (mHAQ) at Day 180 and Day 360
Description: A shortened version of the Health Assessment Questionnaire (HAQ), which uses only 8 instead of the 20 original items and is used to assess motor performance in everyday activities, such as dressing, turning a faucet on/off, and getting in and out of a car. Percent change from baseline = (baseline - post baseline value) / baseline value x 100.
Time Frame: Baseline, Day 180, Day 360
Population: as for outcome 9
Measure: Mean (Standard Error); unit: Percentage of Change on mHAQ scale
Arm/Group | Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) | Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate | Double-Blind (DB) Placebo + Methotrexate
Number analyzed (Participants) | 115 | 105 | 119
Percentage of Change on mHAQ scale
  Mean Percentage Change at Day 180 (n=107, 98, 110) | 41.39 (5.43) | 21.41 (5.67) | 13.73 (5.35)
  Mean PercentageChange at Day 360 (n=109, 100, 111) | 42.49 (5.05) | 22.74 (5.27) | 10.26 (5.00)
Statistical Analysis 1: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Day 180; Test type: Superiority or Other; p = 0.0003, ANCOVA; ANCOVA: % change = pretreatment; Mean Difference (Final Values) = 27.66, 95% CI 2-sided [12.67 to 42.66] — Estimate = adjusted % change (BMS10mg/kg+MTX or BMS 2mg/kg+MTX) - adjusted change for placebo+MTX
Statistical Analysis 2: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Day 180; Test type: Superiority or Other; p = 0.3253, ANCOVA; ANCOVA model: % change = pretreatment; Mean Difference (Final Values) = 7.68 — Estimate = adjusted % change (BMS10mg/kg+MTX or BMS 2mg/kg+MTX) - adjusted change for placebo+MTX
Statistical Analysis 3: Comparison: Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) vs Double-Blind (DB) Placebo + Methotrexate; Day 360; Test type: Superiority or Other; p = 0.0001, ANCOVA; ANCOVA model: % change = pretreatment; Mean Difference (Final Values) = 32.24, 95% CI 2-sided [16.14 to 48.33] — Estimate = adjusted % change (BMS10mg/kg+MTX or BMS 2mg/kg+MTX) - adjusted change for placebo+MTX
Statistical Analysis 4: Comparison: Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate vs Double-Blind (DB) Placebo + Methotrexate; Day 360; Test type: Superiority or Other; p = 0.0869, ANCOVA; ANCOVA model: % change = pretreatment; Mean Difference (Final Values) = 12.48, 95% CI 2-sided [-1.82 to 26.78] — Estimate = adjusted % change (BMS10mg/kg+MTX or BMS 2mg/kg+MTX) - adjusted change for placebo+MTX

11. Secondary Outcome: Number of Participants With At Least One New Active Joint (Tender Joints and Swollen Joints) at Day 180 and Day 360
Time Frame: Day 180, Day 360
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) | Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate | Double-Blind (DB) Placebo + Methotrexate
Number analyzed (Participants) | 115 | 105 | 119
participants
  New Tender Joints(s) at Day 180 | 47 | 65 | 70
  New Swollen Joints(s) at Day 180 | 55 | 59 | 75
  New Tender Joints(s) at Day 360 | 33 | 62 | 69
  New Swollen Joints(s) at Day 360 | 45 | 59 | 69

12. Secondary Outcome: Participants Who Experienced Death, Adverse Events (AEs), Serious AEs (SAEs), and Discontinuations During the Double-Blind Period
Description: AE: any new untoward medical occurrence/worsening of pre-existing medical condition, whether or not related to study drug. SAE: any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; or was an overdose. Participants who discontinued the study due to any AEs were recorded. Related events include those that were considered by the investigator to be certain, probable, or possibly related to study drug.
Time Frame: From the start of study through the end of the double-blind period (at 12 months)
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) | Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate | Double-Blind (DB) Placebo + Methotrexate
Number analyzed (Participants) | 115 | 105 | 119
Participants
  Deaths | 0 | 1 | 0
  SAEs | 14 | 19 | 19
  Discontinuations due to SAEs | 3 | 6 | 3
  Related SAEs | 2 | 5 | 2
  Discontinuations due to AEs | 6 | 10 | 11
  AEs | 104 | 104 | 112
  Related AEs | 56 | 50 | 58

13. Secondary Outcome: Participants With Laboratory Abnormalities Meeting the Marked Abnormality Criteria for Selected Blood Chemistry Values During Double-Blind Therapy
Time Frame: From the start of study up to 60 days post the end of the 12-month double-blind period
Population: Number of Participants Analyzed=All treated participants. n=number of participants evaluated for given measurement.
Measure: Number; unit: Participants
Arm/Group | Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) | Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate | Double-Blind (DB) Placebo + Methotrexate
Number analyzed (Participants) | 115 | 105 | 119
Participants
  High Alanine Aminotransferase (ALT) | 0 | 1 | 2
  High Aspartate Aminotransferase (AST) | 0 | 1 | 0
  High Creatinine | 4 | 3 | 4
  Low Potassium | 2 | 3 | 1
  High Potassium | 1 | 3 | 4

14. Primary Outcome: Participants Receiving Concomitant Disease Modifying Rheumatic Drugs and Biologics in Open-Label (OL) Period
Description: The number of participants receiving concomitant rheumatoid arthritis treatment with disease modifying rheumatic drugs and/or biologics.
Time Frame: Day 360 to Day 3,060
Population: All treated participants.
Measure: Number; unit: Participants
Groups:
- OL Abatacept: Original 10 mg / kg Group: Participants in the double-blind period received a weight-tiered dose of 10 mg/kg of abatacept that was administered monthly by IV infusion over approximately 30 minutes. Participants weighing < 60 kg received abatacept 500 mg, participants weighing ≥ 60 kg and ≤ 100 kg received abatacept 750 mg, and participants > 100 kg received abatacept 1 g. Participants in the present study received an open-label weight-tiered dose of abatacept 10 mg/kg.
- OL Abatacept: Original 2 mg / kg Group: Participants in the double-blind period received a weight-tiered dose of 2 mg/kg of abatacept that was administered monthly by IV infusion over approximately 30 minutes. Participants in the present study received an open-label weight-tiered dose of abatacept 10 mg/kg.
- OL Abatacept: Original Placebo Group: Participants in the double-blind period received a placebo that was administered monthly by IV infusion over approximately 30 minutes. Participants in the present study received an open-label weight-tiered dose of abatacept 10 mg/kg.
Arm/Group | OL Abatacept: Original 10 mg / kg Group | OL Abatacept: Original 2 mg / kg Group | OL Abatacept: Original Placebo Group
Number analyzed (Participants) | 84 | 68 | 67
Participants
  Methotrexate | 84 | 68 | 67
  Corticosteroids (oral and/or injectable) | 72 | 57 | 56
  Nonsteroidal antiinfllammatory drugs | 78 | 63 | 64
  Azanthioprine | 1 | 0 | 1
  Chloroquine | 0 | 1 | 1
  Cyclosporine | 2 | 1 | 0
  Gold Sodium Thiomalate | 0 | 1 | 0
  Hydroxychloroquine | 2 | 3 | 2
  Leflunamide | 2 | 0 | 1
  Sulfasalazine | 0 | 0 | 1
  Adalimumab | 0 | 1 | 0
  Etanercept | 0 | 1 | 0
  Infliximab | 2 | 1 | 0

15. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs) and Serious Adverse Events (SAEs) in OL Period
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with treatment.SAE=any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in development of drug dependency or drug abuse, is an important medical event. Related AE/SAE=Certain,Probable,Possible,or Missing relationship to drug.
Time Frame: Day 360 to Day 3060
Population: All treated OL participants.
Measure: Number; unit: Participants
Groups:
- OL Abatacept (10 mg / kg): OL participants received a weight-tiered dose of 10 mg/kg of abatacept that was administered monthly by an intravenous (IV) infusion over approximately 30 minutes. Participants weighing < 60 kg received abatacept 500 mg, participants weighing ≥ 60 kg and ≤ 100 kg received abatacept 750 mg, and participants > 100 kg received abatacept 1 g.
Arm/Group | OL Abatacept (10 mg / kg)
Number analyzed (Participants) | 219
Participants
  AEs | 211
  Related AEs | 144
  Discontinued Due to AEs | 44
  SAEs | 117
  Related SAEs | 37
  Discontinued Due to SAEs | 33
  Deaths | 8

16. Primary Outcome: Number of Participants With AEs of Special Interest in OL Period
Description: AEs were defined as any new untoward medical occurrence or worsening of a pre- existing medical condition which does not necessarily have a causal relationship with this treatment. AEs of special interest were those which may be associated with the use of immunomodulatory agents or infusion of therapeutic proteins. Acute infusional AEs were defined as those that occurred within 1 hour after the start of the infusion. Peri-Infusional AEs were defined as those that occurred within 24 hours after the start of the infusion.
Time Frame: Day 360 to Day 3060
Population: All treated OL participants.
Measure: Number; unit: Participants
Arm/Group | OL Abatacept (10 mg / kg)
Number analyzed (Participants) | 219
Participants
  Infections/Infestations | 179
  Malignant Neoplasms | 20
  Autoimmune Disorders | 20
  Acute Infusional AEs | 20
  Peri-Infusional AEs | 47

17. Primary Outcome: Baseline Serum Immunoglobulin A (IgA) Over Time in OL Period
Description: Time-matched baseline (Day 0) values and post-baseline values were presented for each post-baseline visit and represent only that cohort of participants with measurements available at that post-baseline assessment. Mean Change from Baseline data for these cohorts are presented in Outcome Measure 6.
Time Frame: Baseline (Day 0) and Days 360, 720,1080, 1440, and 1800
Population: All treated OL participants. Participants were grouped according to the treatment they received in DB study. n=the number of participants with measurements for that time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | OL Abatacept: Original 10 mg / kg Group | OL Abatacept: Original 2 mg / kg Group | OL Abatacept: Original Placebo Group
Number analyzed (Participants) | 84 | 68 | 67
mg/dL
  Baseline for Day 360 cohort (n=74, 59, 60) | 308.09 (152.27) | 341.54 (148.48) | 264.22 (133.90)
  Baseline for Day 720 cohort (n=71, 53, 53) | 290.25 (146.27) | 338.58 (151.76) | 256.64 (132.78)
  Baseline for Day 1080 cohort (n=59, 45, 45) | 287.27 (140.22) | 321.02 (153.81) | 266.89 (143.48)
  Baseline for Day 1440 cohort (n=54, 37, 37) | 287.09 (136.50) | 327.27 (162.13) | 250.11 (127.88)
  Baseline for Day 1800 cohort (n=50, 38, 34) | 292.78 (146.91) | 327.34 (163.27) | 244.71 (118.03)

18. Primary Outcome: Mean Change From Baseline (BL) in IgA Over Time in OL Period
Description: Blood samples for immunoglobulin assessments were obtained to determine change from baseline in serum IgA. Baseline data for these time-matched cohorts are presented in Outcome Measure 5.
Time Frame: Baseline (Day 0) and Days 360, 720, 1080, 1440, and 1800
Population: All treated OL participants. Participants were grouped according to the treatment they received in the DB study. n=the number of participants with measurements for that time point.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | OL Abatacept: Original 10 mg / kg Group | OL Abatacept: Original 2 mg / kg Group | OL Abatacept: Original Placebo Group
Number analyzed (Participants) | 84 | 68 | 67
mg/dL
  Change from BL at Day 360 (n=74, 59, 60) | -38.24 (5.95) | -25.66 (7.83) | 5.00 (6.72)
  Change from BL at Day 720 (n=71, 53, 53) | -28.20 (8.61) | -45.06 (9.27) | -20.89 (7.73)
  Change from BL at Day 1080 (n=59, 45, 45) | -33.10 (13.08) | -52.87 (12.86) | -15.87 (11.18)
  Change from BL at Day 1440 (n=54, 37, 37) | -30.52 (9.75) | -52.49 (16.32) | -4.41 (12.28)
  Change from BL at Day 1800 (n=50, 38, 34) | -20.06 (26.97) | -65.95 (16.26) | -25.68 (12.18)

19. Secondary Outcome: Participants With Laboratory Abnormalities Meeting the Marked Abnormality Criteria for Selected Hematologic Values During Double-Blind Therapy
Time Frame: From the start of study up to 60 days post the end of the 12-month double-blind period
Population: Number of Participants Analyzed=All treated participants. n=number of participants evaluated for given measurement.
Measure: Number; unit: Participants
Arm/Group | Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) | Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate | Double-Blind (DB) Placebo + Methotrexate
Number analyzed (Participants) | 115 | 105 | 119
Participants
  Low Hemoglobin (n=115, 104, 119) | 1 | 0 | 3
  Low Platelets (n=114, 104, 119) | 0 | 0 | 0
  High Platelets (n=114, 104, 119) | 0 | 0 | 0
  Low Leukocytes (n=115, 104, 119) | 0 | 0 | 0
  High Leukocytes (n=115, 104, 119) | 12 | 6 | 14
  Low Neutrophils (n=115, 105, 119) | 0 | 1 | 0

20. Secondary Outcome: Number of Participants Who Discontinued Due to Lack of Efficacy in the DB and OL Periods
Time Frame: Day 1 to Day 360 (Double-Blind Period), Day 361 to Day 3060 (Open-Label Period)
Population: Treated Participants
Measure: Number; unit: participants
Arm/Group | Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) | Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate | Double-Blind (DB) Placebo + Methotrexate | Open-Label (OL) Abatacept (10 mg / kg)
Number analyzed (Participants) | 115 | 105 | 119 | 219
participants | 12 | 16 | 28 | 26

21. Secondary Outcome: Immunogenicity Data: Anti-CTLA4Ig Antibodies With Immunoglobulin (IG) Region
Time Frame: Baseline, Days 30, 90, 180, 270, 360
Population: Number of Participants Analyzed=treated participants; n=number of participants with both baseline and post-baseline measurements at timepoint.
Measure: Geometric Mean (Standard Deviation); unit: titers
Arm/Group | Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) | Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate
Number analyzed (Participants) | 115 | 105
titers
  Baseline for Day 30 Cohort (n=110, 100) | 9151.8 (10692.68) | 8861.8 (9282.06)
  Day 30 (n=110, 100) | 8361.5 (9931.79) | 8561.7 (9323.91)
  Baseline for Day 90 Cohort (n=110, 99) | 9052.8 (10392.26) | 8930.2 (9002.57)
  Day 90 (n=110, 99) | 6842.3 (7659.01) | 7497.8 (7356.42)
  Baseline for Day 180 Cohort (n=102, 90) | 8853.6 (10330.92) | 8689.3 (8626.90)
  Day 180 (n=102, 90) | 5967.3 (6535.57) | 7016.5 (6945.59)
  Baseline for Day 270 Cohort (n=94, 73) | 13149.7 (14850.07) | 11976.7 (13679.48)
  Day 270 (n=94, 73) | 8027.5 (8863.47) | 9725.9 (11337.20)
  Baseline for Day 360 Cohort (n=83, 74) | 13287.8 (15024.78) | 11712.4 (12971.16)
  Day 360 (n=83, 74) | 8675.1 (10038.76) | 10284.1 (12175.48)

22. Secondary Outcome: Immunogenicity Data: Anti-CTLA4Ig Antibodies Without IG Region
Time Frame: Baseline, Days 30, 90, 180, 270, 360
Population: as for outcome 21
Measure: Geometric Mean (Standard Deviation); unit: titers
Arm/Group | Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) | Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate
Number analyzed (Participants) | 115 | 105
titers
  Baseline for Day 30 Cohort (n=110, 101) | 12.6 (9.59) | 11.7 (4.79)
  Day 30 (n=110, 101) | 12.5 (9.38) | 12.0 (5.58)
  Baseline for Day 90 Cohort (n=110, 99) | 12.5 (9.42) | 11.6 (4.69)
  Day 90 (n=110, 99) | 12.0 (8.31) | 11.4 (3.96)
  Baseline for Day 180 Cohort (n=102, 90) | 12.6 (9.91) | 11.6 (4.76)
  Day 180 (n=102, 90) | 12.1 (8.66) | 11.7 (5.01)
  Baseline for Day 270 Cohort (n=95, 73) | 13.4 (10.51) | 12.1 (5.22)
  Day 270 (n=95, 73) | 12.5 (8.70) | 11.7 (4.42)
  Baseline for Day 360 Cohort (n=84, 76) | 13.6 (11.03) | 12.2 (5.77)
  Day 360 (n=84, 76) | 12.9 (9.79) | 11.6 (4.42)

23. Secondary Outcome: Immunogenicity Data: Categories of Post Baseline Value to Baseline Value (VA/PRE) Ratios and Number of Participants With Sero-conversion (Anti-CTLA4Ig Antibodies With IG Region)
Description: Number of participants with ratio of VA/PRE <=3, <3 to <=9, and >9. Ratios greater than 9 are incidences of Anti-CTLA4Ig sero-conversion.
Time Frame: Baseline, Days 30, 90, 180, 270, 360
Population: as for outcome 21
Measure: Number; unit: participants
Arm/Group | Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) | Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate
Number analyzed (Participants) | 115 | 105
participants
  Day 30, ratio <=3 (n=110, 100) | 109 | 100
  Day 30, ratio <3 to <=9 (n=110, 100) | 1 | 0
  Day 30, ratio >9 (n=110, 100) | 0 | 0
  Day 90, ratio <=3 (n=110, 99) | 110 | 99
  Day 90, ratio <3 to <=9 (n=110, 99) | 0 | 0
  Day 90, ratio >9 (n=110, 99) | 0 | 0
  Day 180, ratio <=3 (n=102, 90) | 101 | 90
  Day 180, ratio <3 to <=9 (n=102, 90) | 1 | 0
  Day 180, ratio >9 (n=102, 90) | 0 | 0
  Day 270, ratio <=3 (n=94, 73) | 94 | 73
  Day 270, ratio <3 to <=9 (n=94, 73) | 0 | 0
  Day 270, ratio >9 (n=94, 73) | 0 | 0
  Day 360, ratio <=3 (n=83, 74) | 81 | 72
  Day 360, ratio <3 to <=9 (n=83, 74) | 2 | 2
  Day 360, ratio >9 (n=83, 74) | 0 | 0

24. Primary Outcome: Baseline Immunoglobulin G (IgG) Over Time in OL Period
Description: Time-matched baseline (Day 0) values and post-baseline vales were presented for each post-baseline visit and represent only that cohort of participants with measurements available at that post-baseline assessment. Mean Change from Baseline data for these cohorts are presented in Outcome Measure 8.
Time Frame: Baseline (Day 0) and Days 360, 720, 1080, 1440 and 1800
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- OL Abatacept: Original 10 mg / kg Group: Participants in the DB period received a weight-tiered dose of 10 mg/kg of abatacept that was administered monthly by IV infusion over approximately 30 minutes. Participants weighing < 60 kg received abatacept 500 mg, participants weighing ≥ 60 kg and ≤ 100 kg received abatacept 750 mg, and participants > 100 kg received abatacept 1 g. Participants in the present study received an OL weight-tiered dose of abatacept 10 mg/kg.
- OL Abatacept: Original 2 mg / kg Group: Participants in the DB period received a weight-tiered dose of 2 mg/kg of abatacept that was administered monthly by IV infusion over approximately 30 minutes. Participants in the present study received an OL weight-tiered dose of abatacept 10 mg/kg.
Arm/Group | OL Abatacept: Original 10 mg / kg Group | OL Abatacept: Original 2 mg / kg Group | OL Abatacept: Original Placebo Group
Number analyzed (Participants) | 84 | 68 | 67
mg/dL
  Baseline for Day 360 cohort (n=75, 59, 60) | 1130.31 (295.28) | 1086.05 (263.41) | 1079.00 (345.72)
  Baseline for Day 720 cohort (n=72, 53, 53) | 1138.58 (303.24) | 1093.23 (318.24) | 1076.40 (333.08)
  Baseline for Day 1080 cohort (n=60, 45, 45) | 1145.15 (305.51) | 1053.91 (264.53) | 1136.27 (372.58)
  Baseline for Day 1440 cohort (n=55, 37, 37) | 1154.58 (315.00) | 1095.49 (261.86) | 1135.43 (381.72)
  Baseline for Day 1800 cohort (n=51, 38, 34) | 1152.63 (305.01) | 1092.76 (260.85) | 1137.21 (368.39)

25. Primary Outcome: Mean Change From Baseline (BL) in IgG Over Time in OL Period
Description: Blood samples for immunoglobulin assessments were obtained to determine change from baseline in serum IgG. Baseline data for these cohorts are presented in Outcome Measure 7.
Time Frame: Baseline (Day 0) and Days 360, 720, 1080, 1440, and 1800
Population: as for outcome 18
Measure: Mean (Standard Error); unit: mg/dL
Groups:
- OL Abatacept: Original Placebo Group: Participants in the DB period received a placebo that was administered monthly by IV infusion over approximately 30 minutes. Participants in the present study received an OL weight-tiered dose of abatacept 10 mg/kg.
Arm/Group | OL Abatacept: Original 10 mg / kg Group | OL Abatacept: Original 2 mg / kg Group | OL Abatacept: Original Placebo Group
Number analyzed (Participants) | 84 | 68 | 67
mg/dL
  Change from BL at Day 360 (n=75, 59, 60) | -181.92 (19.78) | -110.71 (21.46) | -15.12 (21.71)
  Change from BL at Day 720 (n=72, 53, 53) | -183.04 (28.58) | -168.55 (31.82) | -137.06 (31.62)
  Change from BL at Day 1080 (n=60, 45, 45) | -199.58 (33.68) | -229.91 (26.75) | -150.40 (33.97)
  Change from BL at Day 1440 (n=55, 37, 37) | -228.11 (28.90) | -279.14 (33.43) | -147.46 (45.84)
  Change from BL at Day 1800 (n=51, 38, 34) | -217.43 (39.52) | -206.21 (39.10) | -187.94 (44.40)

26. Primary Outcome: Baseline Immunoglobulin M (IgM) Over Time in OL Period
Description: Time-matched baseline (Day 0) values and post-baseline values were presented for each post-baseline visit and represent only that cohort of participants with measurements available at that post-baseline assessment. Mean Change from Baseline data for these cohorts are presented in Outcome Measure 10.
Time Frame: Baseline (Day 0) and Days 360, 720,1080,1440, and 1800
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | OL Abatacept: Original 10 mg / kg Group | OL Abatacept: Original 2 mg / kg Group | OL Abatacept: Original Placebo Group
Number analyzed (Participants) | 84 | 68 | 67
mg/dL
  Baseline for Day 360 cohort (n=74, 59, 60) | 147.76 (76.05) | 134.29 (66.81) | 125.10 (52.12)
  Baseline for Day 720 cohort (n=71, 53, 53) | 147.76 (76.31) | 137.79 (69.93) | 123.25 (52.79)
  Baseline for Day 1080 cohort (n=59, 45, 45) | 144.75 (78.89) | 127.36 (68.06) | 129.04 (54.79)
  Baseline for Day 1440 cohort (n=54, 37, 37) | 141.69 (77.90) | 136.22 (70.90) | 133.51 (58.04)
  Baseline for Day 1800 cohort (n=45, 33, 32) | 133.22 (61.79) | 124.15 (67.07) | 124.63 (58.69)

27. Secondary Outcome: Immunogenicity Data: Categories of Post Baseline Value to Baseline Value (VA/PRE) Ratios and Number of Participants With Sero-conversion(Anti-CTLA4Ig Antibodies Without IG Region)
Description: as for outcome 23
Time Frame: Baseline, Days 30, 90, 180, 270, 360
Population: as for outcome 21
Measure: Number; unit: participants
Arm/Group | Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) | Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate
Number analyzed (Participants) | 115 | 105
participants
  Day 30, ratio <=3 (n=110, 101) | 108 | 99
  Day 30, ratio <3 to <=9 (n=110, 101) | 1 | 2
  Day 30, ratio >9 (n=110, 101) | 1 | 0
  Day 90, ratio <=3 (n=110, 99) | 110 | 99
  Day 90, ratio <3 to <=9 (n=110, 99) | 0 | 0
  Day 90, ratio >9 (n=110, 99) | 0 | 0
  Day 180, ratio <=3 (n=102, 90) | 101 | 89
  Day 180, ratio <3 to <=9 (n=102, 90) | 1 | 0
  Day 180, ratio >9 (n=102, 90) | 0 | 1
  Day 270, ratio <=3 (n=95, 73) | 95 | 73
  Day 270, ratio <3 to <=9 (n=95, 73) | 0 | 0
  Day 270, ratio >9 (n=95, 73) | 0 | 0
  Day 360, ratio <=3 (n=84, 76) | 84 | 76
  Day 360, ratio <3 to <=9 (n=84, 76) | 0 | 0
  Day 360, ratio >9 (n=84, 76) | 0 | 0

28. Secondary Outcome: Pharmacodynamic Measure: Mean Changes From Baseline in Rheumatoid Factor at Day 180 and Day 360
Time Frame: Baseline, Day 180, Day 360
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) | Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate | Double-Blind (DB) Placebo + Methotrexate
Number analyzed (Participants) | 115 | 105 | 119
IU/mL
  Mean Change at Day 180 (n=95, 84, 74) | -104.3 [-151.5 to 57.0] | -28.1 [-52.1 to -4.1] | -0.6 [-31.7 to 30.4]
  Mean Change at Day 360 (n=69, 54, 57) | -118.3 [-175.2 to -61.4] | -23.6 [-56.8 to 9.7] | 20.9 [-11.3 to 53.1]

29. Secondary Outcome: Pharmacodynamic Measure: Mean Changes From Baseline in Interleukin-6 at Day 180 and Day 360
Time Frame: Baseline, Day 180, Day 360
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) | Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate | Double-Blind (DB) Placebo + Methotrexate
Number analyzed (Participants) | 115 | 105 | 119
pg/mL
  Mean Change at Day 180 (n=85, 74, 68) | -20.5 [-27.8 to -13.2] | -16.1 [-24.2 to -8.0] | 1.3 [-7.9 to 10.5]
  Mean Change at Day 360 (n=56, 47, 47) | -20.9 [-31.6 to -10.2] | -12.7 [-22.5 to -2.9] | -0.6 [-8.1 to 6.9]

30. Secondary Outcome: Pharmacodynamic Measure: Mean Changes From Baseline in Plasma Soluble Interleukin-2 Receptor (sIL-2R) at Day 180 and Day 360
Time Frame: Baseline, Day 180, Day 360
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) | Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate | Double-Blind (DB) Placebo + Methotrexate
Number analyzed (Participants) | 115 | 105 | 119
pg/mL
  Mean Change at Day 180 (n=94, 84, 76) | -315.9 [-418.5 to -213.3] | -135.5 [-241.5 to -29.5] | 43.6 [-71.2 to 158.4]
  Mean Change at Day 360 (n=68, 55, 54) | -194.3 [-305.7 to -83.0] | 40.4 [-71.5 to 152.3] | 196.8 [24.3 to 369.4]

31. Secondary Outcome: Pharmacodynamic Measure: Mean Changes From Baseline in E-Selectin at Day 180 and Day 360
Time Frame: Baseline, Day 180, Day 360
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) | Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate | Double-Blind (DB) Placebo + Methotrexate
Number analyzed (Participants) | 115 | 105 | 119
ng/mL
  Mean Change at Day 180 (n=88, 80, 71) | -8.3 [-13.2 to -3.4] | 0.5 [-6.0 to 7.0] | -0.7 [-6.9 to 5.5]
  Mean Change at Day 360 (n=75, 67, 61) | -10.9 [-15.7 to -6.1] | 0.6 [-6.0 to 9.0] | 2.0 [-4.9 to 9.0]

32. Secondary Outcome: Pharmacodynamic Measure: Mean Changes From Baseline in Soluble Inter-Cellular Adhesion Molecule 1 (sICAM-1) at Day 180 and Day 360
Time Frame: Baseline, Day 180, Day 360
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) | Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate | Double-Blind (DB) Placebo + Methotrexate
Number analyzed (Participants) | 115 | 105 | 119
ng/mL
  Mean Change at Day 180 (n=94, 82, 75) | -40.6 [-58.5 to -22.8] | -6.2 [-27.5 to 15.1] | 1.1 [-31.9 to 34.1]
  Mean Change at Day 360 (n=77, 67, 63) | -55.2 [-74.8 to -35.5] | -13.6 [-36.3 to 9.0] | 0.7 [-27.6 to 28.9]

33. Secondary Outcome: Pharmacodynamic Measure: Mean Changes From Baseline in Tumor Necrosis Factor (TNF)-Alpha at Day 180 and Day 360
Time Frame: Baseline, Day 180, Day 360
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Double-Blind (DB) Abatacept 10 mg/kg + Methotrexate (MTX) | Double-Blind (DB) Abatacept 2 mg/kg + Methotrexate | Double-Blind (DB) Placebo + Methotrexate
Number analyzed (Participants) | 115 | 105 | 119
ng/mL
  Mean Change at Day 180 (n=83, 74, 68) | -3.7 [-8.7 to 1.3] | -1.2 [-4.3 to 1.9] | -3.6 [-8.0 to 0.7]
  Mean Change at Day 360 (n=61, 48, 49) | -3.0 [-8.7 to 2.7] | 1.1 [-1.3 to 3.4] | -0.3 [-3.2 to 2.7]

34. Secondary Outcome: Number of ACR 20 Responders in OL Period
Description: as for outcome 1
Time Frame: Days 360, 450, 540, 630, 720, 810, 900, 1080, 1350, 1440, 1530, 1620, 1710, 1800, 1980, 2160, 2340, 2520, 2700, 2880, and 3060
Population: All treated OL participants. Participants were grouped according to the treatment they received in the double-blind (DB) study. N = number of participants analyzed and n = the number of participants with measurements for that time point.
Measure: Number; unit: Participants
Groups:
- OL Abatacept: Original 10 mg/kg Group: Participants in the double-blind period received a weight-tiered dose of 10 mg/kg of abatacept that was administered monthly by an intravenous (IV) infusion over approximately 30 minutes. Participants weighing < 60 kg received abatacept 500 mg, participants weighing ≥ 60 kg and ≤ 100 kg received abatacept 750 mg, and participants > 100 kg received abatacept 1 g. Participants in the present study received an open-label weight-tiered dose of abatacept 10 mg/kg.
- OL Abatacept: Original 2 mg/kg Group: Participants in the double-blind period received a weight-tiered dose of 2 mg/kg of abatacept that was administered monthly by an intravenous (IV) infusion over approximately 30 minutes. Participants in the present study received an open-label weight-tiered dose of abatacept 10 mg/kg.
- OL Abatacept: Original Placebo Group: Participants in the double-blind period received a placebo that was administered monthly by an intravenous (IV) infusion over approximately 30 minutes. Participants in the present study received an open-label weight-tiered dose of abatacept 10 mg/kg.
Arm/Group | OL Abatacept: Original 10 mg/kg Group | OL Abatacept: Original 2 mg/kg Group | OL Abatacept: Original Placebo Group
Number analyzed (Participants) | 84 | 68 | 67
Participants
  Day 360 (n=84, 68, 67) | 64 | 40 | 37
  Day 450 (n=83, 67, 66) | 56 | 45 | 46
  Day 540 (n=82, 65, 59) | 61 | 45 | 45
  Day 630 (n=79, 63, 59) | 60 | 44 | 44
  Day 720 (n=75, 59, 56) | 58 | 39 | 43
  Day 810 (n=73, 56, 54) | 49 | 41 | 44
  Day 900 (n=69, 53, 51) | 56 | 42 | 42
  Day 990 (n=66, 52, 51) | 52 | 39 | 40
  Day 1080 (n=66, 50, 49) | 48 | 39 | 35
  Day 1170 (n=65, 50, 49) | 46 | 35 | 36
  Day 1260 (n=64, 49, 46) | 48 | 41 | 39
  Day 1350 (n=62, 48, 44) | 46 | 30 | 37
  Day 440 (n=61, 47, 44) | 43 | 38 | 37
  Day 1530 (n=60, 46, 43) | 45 | 35 | 29
  Day 1620 (n=58, 45, 43) | 44 | 35 | 38
  Day 1710 (n=58, 45, 42) | 37 | 34 | 38
  Day 1800 (n=56, 44, 42) | 44 | 32 | 38
  Day 1980 (n=53, 44, 40) | 37 | 34 | 28
  Day 2160 (n=49, 42, 38) | 39 | 33 | 32
  Day 2340 (n=47, 36, 36) | 35 | 27 | 28
  Day 2520 (n=43, 37, 33) | 31 | 30 | 28
  Day 2700 (n=37, 34, 34) | 33 | 26 | 23
  Day 2880 (n=36, 31, 32) | 28 | 28 | 27
  Day 3060 (n=18, 18, 17) | 13 | 13 | 14

35. Secondary Outcome: Number of ACR 50 Responders in the OL Period
Description: as for outcome 3
Time Frame: as for outcome 34
Population: All treated OL participants. Participants were grouped according to the treatment they received in the DB study. N=number of participants analyzed; n=the number of participants with measurements for that time point.
Measure: Number; unit: Participants
Groups:
- OL Abatacept: Original 10 mg/kg Group: Participants in the DBperiod received a weight-tiered dose of 10 mg/kg of abatacept that was administered monthly by IV infusion over approximately 30 minutes. Participants weighing <60 kg received abatacept 500 mg, participants weighing ≥60 kg and ≤100 kg received abatacept 750 mg, and participants >100 kg received abatacept 1 g. Participants in the present study received an OL weight-tiered dose of abatacept 10 mg/kg.
- OL Abatacept: Original 2 mg/kg Group: Participants in the DB period received a weight-tiered dose of 2 mg/kg of abatacept that was administered monthly by IV infusion over approximately 30 minutes. Participants in the present study received an OL weight-tiered dose of abatacept 10 mg/kg.
Arm/Group | OL Abatacept: Original 10 mg/kg Group | OL Abatacept: Original 2 mg/kg Group | OL Abatacept: Original Placebo Group
Number analyzed (Participants) | 84 | 68 | 67
Participants
  Day 360 (n=84, 68, 67) | 44 | 23 | 21
  Day 450 (n=83, 67, 66) | 41 | 30 | 30
  Day 540 (n=82, 65, 59) | 38 | 28 | 31
  Day 630 (n=79, 63, 59) | 38 | 27 | 31
  Day 720 (n=75, 59, 56) | 43 | 29 | 34
  Day 810 (n=73, 56, 54) | 42 | 23 | 30
  Day 900 (n=69, 53, 51) | 40 | 34 | 29
  Day 990 (n=66, 52, 51) | 40 | 28 | 31
  Day 1,080 (n=66, 50, 49) | 35 | 24 | 29
  Day 1,170 (n=65, 50, 49) | 36 | 27 | 29
  Day 1,260 (n=64, 49, 46) | 33 | 24 | 28
  Day 1,350 (n=62, 48, 44) | 28 | 24 | 28
  Day 1,440 (n=61, 47, 44) | 25 | 33 | 24
  Day 1,530 (n=60, 46, 43) | 33 | 28 | 26
  Day 1,620 (n=58, 45, 43) | 29 | 27 | 26
  Day 1,710 (n=58, 45, 42) | 23 | 27 | 25
  Day 1,800 (n=56, 44, 42) | 34 | 28 | 28
  Day 1,980 (n=53, 44, 40) | 31 | 26 | 22
  Day 2,160 (n=49, 42, 38) | 25 | 30 | 25
  Day 2,340 (n=47, 36, 36) | 24 | 15 | 21
  Day 2,520 (n=43, 37, 33) | 25 | 23 | 21
  Day 2,700 (n=37, 34, 34) | 23 | 19 | 17
  Day 2,880 (n=36, 31, 32) | 23 | 18 | 19
  Day 3,060 (n=18, 18, 17) | 8 | 10 | 9

36. Secondary Outcome: Number of ACR 70 Responders in the OL Period
Description: ACR 70 response requires a participant to have a 70% reduction in the number of swollen and tender joints, and a reduction of 70% in 3 of the following 5 parameters: physician global assessment of disease, participant global assessment of disease, participant assessment of pain, C-reactive protein or erythrocyte sedimentation rate, and degree of disability in HAQ score. A participant achieved a sustained ACR 70 response if the participant had ACR 70 observed for at least 2 consecutive study visits.
Time Frame: as for outcome 34
Population: as for outcome 35
Measure: Number; unit: Participants
Groups:
- OL Abatacept: Original 10 mg/kg: Participants in the DB period received a weight-tiered dose of 10 mg/kg of abatacept that was administered monthly by IV infusion over approximately 30 minutes. Participants weighing <60 kg received abatacept 500 mg, participants weighing ≥60 kg and ≤100 kg received abatacept 750 mg, and participants >100 kg received abatacept 1 g. Participants in the present study received an OL weight-tiered dose of abatacept 10 mg/kg.
- OL Abatacept: Original 2 mg/kg: Participants in the DB period received a weight-tiered dose of 2 mg/kg of abatacept that was administered monthly by IV infusion over approximately 30 minutes. Participants in the present study received an OL weight-tiered dose of abatacept 10 mg/kg.
- OL Abatacept: Original Placebo: Participants in the DB period received a placebo that was administered monthly by IV infusion over approximately 30 minutes. Participants in the present study received an OL weight-tiered dose of abatacept 10 mg/kg.
Arm/Group | OL Abatacept: Original 10 mg/kg | OL Abatacept: Original 2 mg/kg | OL Abatacept: Original Placebo
Number analyzed (Participants) | 84 | 68 | 67
Participants
  Day 360 (n=84, 68, 67) | 24 | 13 | 9
  Day 450 (n=83, 67, 66) | 21 | 14 | 12
  Day 540 (n=82, 65, 59) | 28 | 15 | 12
  Day 630 (n=79, 63, 59) | 25 | 17 | 15
  Day 720 (n=75, 59, 56) | 22 | 18 | 16
  Day 810 (n=73, 56, 54) | 20 | 14 | 11
  Day 900 (n=69, 53, 51) | 19 | 16 | 15
  Day 990 (n=66, 52, 51) | 23 | 17 | 17
  Day 1080 (n=66, 50, 49) | 21 | 18 | 16
  Day 1170 (n=65, 50, 49) | 23 | 16 | 17
  Day 1260 (n=64, 49, 46) | 20 | 12 | 20
  Day 1350 (n=62, 48, 44) | 18 | 13 | 13
  Day 1440 (n=61, 47, 44) | 19 | 16 | 15
  Day 1530 (n=60, 46, 43) | 22 | 16 | 13
  Day 1620 (n=58, 45, 43) | 21 | 15 | 16
  Day 1710 (n=58, 45, 42) | 15 | 18 | 12
  Day 1800 (n=56, 44, 42) | 21 | 17 | 15
  Day 1980 (n=53, 44, 40) | 25 | 16 | 10
  Day 2160 (n=49, 42, 38) | 23 | 18 | 11
  Day 2340 (n=47, 36, 36) | 19 | 11 | 14
  Day 2520 (n=43, 37, 33) | 19 | 16 | 11
  Day 2700 (n=37, 34, 34) | 20 | 12 | 12
  Day 2880 (n=36, 31, 32) | 17 | 10 | 12
  Day 3060 (n=18, 18, 17) | 6 | 6 | 7

37. Secondary Outcome: Number of Participants With a Clinically Meaningful Improvement on the Modified Health Assessment Questionnaire (mHAQ) in OL Period
Description: The mHAQ is a self-administered questionnaire composed of 20 questions that assess physical functions in 8 domains: dressing, arising, eating, walking, hygiene, reach, grip, and common activities. The answers are graded on a 4-point scale: 0=without any difficulty, 1=with some difficulty, 2=with much difficulty, and 3=unable to do. The HAQ disease index is a weighted sum of the scale scores, with a higher score indicating poorer function. A clinically meaningful improvement was defined as a reduction from baseline in mHAQ score of at least 0.30 units.
Time Frame: Days 360, 720,1080, 1440, 1800, 2160, 2520, 2880, and 3060
Population: All treated OL participants. Participants were grouped according to the treatment they received in the DB study. N =number of participants analyzed; n=the number of participants with measurements for that time point.
Measure: Number; unit: Participants
Groups:
- OL Abatacept: Original Placebo: Participants in the DB period received a placebo that was administered monthly by IV infusion over approximately 30 minutes. Participants in the present study received an on OL weight-tiered dose of abatacept 10 mg/kg.
Arm/Group | OL Abatacept: Original 10 mg/kg | OL Abatacept: Original 2 mg/kg | OL Abatacept: Original Placebo
Number analyzed (Participants) | 84 | 68 | 67
Participants
  Day 360 (n=84, 68, 67) | 46 | 30 | 23
  Day 720 (n=75, 59, 56) | 39 | 34 | 21
  Day 1080 (n=66, 50, 49) | 34 | 28 | 28
  Day 1440 (n=61, 47, 44) | 31 | 26 | 20
  Day 1800 (n=56, 44, 42) | 29 | 27 | 20
  Day 2160 (n=49, 42, 38) | 26 | 24 | 15
  Day 2520 (n=43, 37, 33) | 23 | 21 | 17
  Day 2880 (n=36, 31, 32) | 18 | 21 | 14
  Day 3060 (n=18, 18, 17) | 8 | 8 | 5

38. Secondary Outcome: Baseline Level of Serum Rheumatoid Factor Over Time in OL Period
Description: Serum evaluations were carried out to determine participant baseline rheumatoid factor serum concentration. Time-matched baseline(Day 0) values and post-baseline vales were presented for each post-baseline visit and represent only that cohort of participants with measurements available at that post-baseline assessment.
Time Frame: Baseline (Day 0) and Days 360, 720,1080, 1440, 1800, 2160, 2520, 2880, and 3060
Population: All treated OL participants. Participants were grouped according to the treatment they received in the DB study. n =the number of participants with measurements for that time point.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | OL Abatacept: Original 10 mg/kg | OL Abatacept: Original 2 mg/kg | OL Abatacept: Original Placebo
Number analyzed (Participants) | 84 | 68 | 67
IU/mL
  Baseline for Day 360 cohort (n=80, 62, 65) | 291.98 (374.41) | 219.24 (262.55) | 233.57 (299.75)
  Baseline for Day 720 cohort (n=69, 57, 54) | 256.12 (361.74) | 217.21 (267.03) | 227.81 (308.53)
  Baseline for Day 1080 cohort (n=64, 49, 47) | 233.95 (346.73) | 172.00 (204.63) | 203.94 (250.44)
  Baseline for Day 1440 cohort (n=57, 41, 41) | 243.32 (363.86) | 165.39 (173.31) | 215.71 (258.60)
  Baseline for Day 1800 cohort (n=51, 41, 40) | 165.39 (152.94) | 175.41 (206.37) | 205.33 (254.25)
  Baseline for Day 2160 (n=43, 34, 30) | 185.74 (173.26) | 181.91 (216.48) | 194.17 (254.30)
  Baseline for Day 2520 (n=23, 24, 22) | 175.13 (156.99) | 158.42 (210.74) | 269.55 (309.15)
  Baseline for Day 2880 (n=15, 16, 13) | 159.93 (123.69) | 197.63 (251.82) | 366.38 (362.39)
  Baseline for Day 3060 (n=7, 9, 5) | 214.29 (120.00) | 223.44 (316.59) | 232.60 (202.38)

39. Secondary Outcome: Mean Change From Baseline in Serum Rheumatoid Factor Level Over Time in OL Period
Description: Serum evaluations were carried out to determine participant change from baseline in rheumatoid factor serum concentration. Mean change from baseline = value at post-baseline OL time point-value and baseline OL time point.
Time Frame: Baseline (Day 0) and Days 360, 720,1080, 1440, 1800, 2160, 2520, 2880, and 3060
Population: as for outcome 38
Measure: Mean (Standard Error); unit: IU/mL
Arm/Group | OL Abatacept: Original 10 mg/kg | OL Abatacept: Original 2 mg/kg | OL Abatacept: Original Placebo
Number analyzed (Participants) | 84 | 68 | 67
IU/mL
  Change at Day 360 (n=80, 62, 65) | -72.78 (39.69) | -21.71 (14.50) | 7.77 (21.05)
  Change at Day 720 (n=69, 57, 54) | 37.51 (76.03) | -40.23 (23.05) | -48.37 (48.47)
  Change at Day 1080 (n=64, 49, 47) | 8.53 (66.71) | -34.78 (24.22) | -0.04 (38.15)
  Change at Day 1440 (n=57, 41, 41) | 43.81 (97.15) | -15.68 (32.26) | 1.54 (49.24)
  Change at Day 1800 (n=51, 41, 40) | 30.29 (30.78) | 10.95 (41.17) | -49.83 (40.58)
  Change at Day 2160 (n=43, 34, 30) | -8.44 (45.19) | -26.29 (35.06) | -65.50 (51.49)
  Change at Day 2520 (n=23, 24, 22) | 87.61 (99.50) | -54.92 (41.93) | -50.05 (70.38)
  Change at Day 2880 (n=15, 16, 13) | 28.47 (45.91) | -102.06 (64.62) | 46.54 (193.55)
  Change at Day 3060 (n=7, 9, 5) | -45.14 (88.72) | -89.00 (109.53) | 118.40 (252.72)

40. Primary Outcome: Mean Change From Baseline (BL) in IgM in OL Period
Description: Blood samples for immunoglobulin assessments were obtained to determine change from baseline in serum IgM. Baseline data for these time-matched cohorts are presented in Outcome Measure 9.
Time Frame: Baseline (Day 0) and Days 360, 720, 1080, 1440, and 1800
Population: All treated OL participants. Participants were grouped according to the treatment they received in the double-blind (DB) study. n = the number of participants with measurements for that time point.
Measure: Mean (Standard Error); unit: mg/dL
Groups:
- OL Abatacept: Original 10 mg/kg Group: Participants in the DB period received a weight-tiered dose of 10 mg/kg of abatacept that was administered monthly by intravenous IV infusion over approximately 30 minutes. Participants weighing < 60 kg received abatacept 500 mg, participants weighing ≥ 60 kg and ≤ 100 kg received abatacept 750 mg, and participants > 100 kg received abatacept 1 g. Participants in the present study received an OL weight-tiered dose of abatacept 10 mg/kg.
Arm/Group | OL Abatacept: Original 10 mg/kg Group | OL Abatacept: Original 2 mg/kg Group | OL Abatacept: Original Placebo Group
Number analyzed (Participants) | 84 | 68 | 67
mg/dL
  Change from BL at Day 360 (n=74, 59, 60) | -5.81 (3.49) | 3.22 (4.36) | 11.17 (3.89)
  Change from BL at Day 720 (n=71, 53, 53) | 12.68 (7.32) | 0.11 (4.76) | 6.45 (6.11)
  Change from BL at Day 1080 (n=59, 45, 45) | 0.37 (6.69) | 1.93 (6.61) | 27.93 (11.62)
  Change from BL at Day 1440 (n=54, 37, 37) | 2.52 (7.07) | 0.68 (8.99) | 14.46 (9.52)
  Change from BL at Day 1,800 (n=45, 33, 32) | 7.84 (6.89) | 9.06 (7.55) | 6.72 (8.80)

41. Primary Outcome: Number of Participants With Hematology Values Meeting Marked Abnormality Criteria in OL Period
Time Frame: Day 360 to Day 3060
Population: All treated OL participants.
Measure: Number; unit: Participants
Groups:
- OL Abatacept (10 mg / kg): OL participants received a weight-tiered dose of 10 mg/kg of abatacept that was administered monthly by IV infusion over approximately 30 minutes. Participants weighing < 60 kg received abatacept 500 mg, participants weighing ≥ 60 kg and ≤ 100 kg received abatacept 750 mg, and participants > 100 kg received abatacept 1 g.
Arm/Group | OL Abatacept (10 mg / kg)
Number analyzed (Participants) | 217
Participants
  Low Hemoglobin (> 13.0 grams/dL; n=216) | 21
  Low Hematocrit (< 35%; n=216) | 11
  Low Platelet Count (<145*10^9 cells/L; n=214) | 1
  High Platelet Count (>400*10^9 cells/L; n=214) | 1
  Low Leukocytes (<3.60 *10^3 cells/µL; n=216) | 12
  High Leukocytes (>10.30*10^3 cells/µL; n=216) | 49
  Low Neutrophils + Bands (<2.0*10^3 c/uL; n=217) | 1
  Low Absolute Lymphocytes(<1.0*10^3cells/µL; n=217) | 48
  High Absolute Lymphocytes(>3.5*10^3cells/µL;n=217) | 0
  High Absolute Monocytes (>720*10^3cells/µL; n=217) | 0
  High Absolute Basophils(>0.2*10^3 cells/µL; n=217) | 1
  High Absolute Eosinophils(>0.4*10^3cells/µL;n=217) | 21

42. Primary Outcome: Number of Participants With Liver and Kidney Function Values Meeting Marked Abnormality Criteria in OL Period
Time Frame: Day 360 to Day 3060
Population: All treated OL participants.
Measure: Number; unit: Participants
Arm/Group | OL Abatacept (10 mg / kg)
Number analyzed (Participants) | 217
Participants
  High Alkaline Phosphatase (>117 IU/L) | 1
  High Aspartate Aminotransferase (>38 IU/L) | 6
  High Alanine Aminotransferase (>30 IU/L) | 5
  High G-Glutamyl Transferase (>61 IU/L) | 20
  High Total Bilirubin (>1.1 mg/dL) | 0
  High Blood Urea Nitrogen (>21.3 mg/dL) | 14
  High Creatinine (>1.30 mg/dL) | 13

43. Primary Outcome: Number of Participants With Electrolyte Values Meeting Marked Abnormality Criteria in OL Period
Time Frame: Day 360 to Day 3060
Population: All treated OL participants.
Measure: Number; unit: Participants
Groups:
- OL Abatacept (10 mg / kg): OL participants received a weight-tiered dose of 10 mg/kg of abatacept that was administered monthly by IV infusion over approximately 30 minutes. Participants weighing <60 kg received abatacept 500 mg, participants weighing ≥60 kg and ≤100 kg received abatacept 750 mg, and participants >100 kg received abatacept 1 g.
Arm/Group | OL Abatacept (10 mg / kg)
Number analyzed (Participants) | 217
Participants
  Low Serum Sodium (<135 mEq/L; n=217) | 4
  High Serum Sodium (>145 mEq/L; n=217) | 10
  Low Serum Potassium (<3.5 mEq/L; n=217) | 8
  High Serum Potassium (>5.0 mEq/L; n=217) | 10
  Low Serum Chloride (<97 mEq/L; n=217) | 8
  High Serum Chloride (>106 mEq/L; n=217) | 3
  Low Total Calcium (<8.6 mg/dL; n=217) | 0
  High Total Calcium (>10.2 mg/dL; n=217) | 3
  Low Inorganic Phosphorus (<2.7 mg/dL; n=217) | 5
  High Inorganic Phosphorus (> 4.5 mg/dL; n=217) | 11

44. Secondary Outcome: Mean Baseline Soluble Serum Interleukin-2 Receptor Level (sIL2-r) Over Time in OL Period
Description: Serum evaluations were carried out to determine participant serum levels of sIL2-r at baseline. Time-matched baseline (Day 0) values and post-baseline vales were presented for each post-baseline visit and represent only that cohort of participants with measurements available at that post-baseline assessment.
Time Frame: Baseline (Day 0) and Days 360, 720,1080, 1440, 1800, 2160, 2520, 2880, and 3060
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- OL Abatacept: Original 10 mg/kg: Participants in the DB period received a weight-tiered dose of 10 mg/kg of abatacept administered monthly by IV infusion over approximately 30 minutes. Participants weighing <60 kg received abatacept 500 mg, participants weighing ≥60 kg and ≤100 kg received abatacept 750 mg, and participants >100 kg received abatacept 1 g. Participants in the present study received an OL weight-tiered dose of abatacept 10 mg/kg.
- OL Abatacept: Original 2 mg /kg: Participants in the DB period received a weight-tiered dose of 2 mg/kg abatacept administered monthly by IV infusion over approximately 30 minutes. Participants in the present study received an OL weight-tiered dose of abatacept 10 mg/kg.
- OL Abatacept: Original Placebo: Participants in the DB period received a placebo administered monthly by IV infusion over approximately 30 minutes. Participants in the present study received an OL weight-tiered dose of abatacept 10 mg/kg.
Arm/Group | OL Abatacept: Original 10 mg/kg | OL Abatacept: Original 2 mg /kg | OL Abatacept: Original Placebo
Number analyzed (Participants) | 84 | 68 | 67
pg/mL
  Baseline for Day 360 cohort (n=69, 57, 58) | 1424.86 (790.75) | 1365.40 (524.90) | 1480.93 (713.88)
  Baseline for Day 720 cohort (n=66, 53, 49) | 1419.82 (721.00) | 1351.15 (497.64) | 1437.24 (730.73)
  Baseline for Day 1080 cohort (n=57, 47, 44) | 1413.28 (760.39) | 1341.51 (520.06) | 1392.09 (678.85)
  Baseline for Day 1440 cohort (n=47, 36, 31) | 1418.64 (806.85) | 1323.14 (538.82) | 1409.71 (687.86)
  Baseline for Day 1800 cohort (n=27, 13, 17) | 1252.04 (572.14) | 1160.15 (444.37) | 1476.06 (590.14)

45. Primary Outcome: Number of Participants With Glucose, Protein, Metabolites, and Urinalysis Values Meeting Marked Abnormality Criteria in OL Period
Time Frame: Day 360 to Day 3060
Population: All treated OL participants.
Measure: Number; unit: Participants
Groups:
- OL Abatacept (10 mg / kg): OL participants received a weight-tiered dose of 10 mg/kg of abatacept that was administered monthly by I) infusion over approximately 30 minutes. Participants weighing <60 kg received abatacept 500 mg, participants weighing ≥60 kg and ≤100 kg received abatacept 750 mg, and participants >100 kg received abatacept 1 g.
Arm/Group | OL Abatacept (10 mg / kg)
Number analyzed (Participants) | 217
Participants
  Low Serum Glucose (< 70 mg/dL; n=217) | 33
  High Serum Glucose (> 110 mg/dL; n=217) | 30
  Low Fasting Serum Glucose (< 70 mg/dL; n=1) | 0
  High Fasting Serum Glucose (> 110 mg/dL; n=1) | 0
  Low Total Protein (< 6.2 grams/dL; n=217) | 12
  High Total Protein (>8.3 grams/dL; n=217) | 1
  Low Albumin (<3.5 grams/dL; n=217) | 7
  High Uric Acid (>7.6 mg/dL; n=217) | 2
  High Urine Protein (> trace; n=217) | 29
  High Urine Glucose (> trace; n=217) | 32
  High Urine Blood (> trace; n=217) | 47
  High Urine White Blood Cell Count (> trace; n=162) | 74
  High Urine Red Blood Cell Count (> trace; n=162) | 51

46. Secondary Outcome: Mean Change From Baseline in sIL2-r Over Time in OL Period
Description: Serum evaluations were carried out to determine participant serum levels of sIL2-r. Mean change from baseline=value at post-baseline OL time point-value and baseline OL time point.
Time Frame: Baseline (Day 0) and Days 360, 720, 1080, 1440, and 1800
Population: as for outcome 38
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | OL Abatacept: Original 10 mg/kg | OL Abatacept: Original 2 mg/kg | OL Abatacept: Original Placebo
Number analyzed (Participants) | 84 | 68 | 67
pg/mL
  Change at Day 360 (n=69, 57, 58) | -200.62 (56.43) | 44.05 (60.80) | 207.40 (91.17)
  Change at Day 720 (n=66, 53, 49) | -323.26 (83.71) | -209.19 (60.08) | -213.22 (83.64)
  Change at Day 1080 (n=57, 47, 44) | -158.93 (96.60) | -44.98 (95.04) | -156.20 (69.04)
  Change at Day 1440 (n=47, 36, 31) | -421.57 (98.79) | -392.08 (81.78) | -394.45 (123.99)
  Change at Day 1800 (n=27, 13, 17) | -249.81 (123.30) | -84.77 (61.61) | -247.12 (128.65)

47. Secondary Outcome: Mean Baseline Serum C-Reactive Protein Level Over Time in OL Period
Description: Serum evaluations were carried out to evaluate participant serum CRP concentrations at baseline. Time-matched BL (Day 0) values and post-BL vales were presented for each post-BL visit and represent only that cohort of participants with measurements available at that post-BL assessment.
Time Frame: Baseline (Day 0) and Days 360, 720, 1080,1440,1800, 2160, 2520, 2880, 3060
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- OL Abatacept: Original 2 mg/kg: Participants in the DB period received a weight-tiered dose of 2 mg/kg of abatacept administered monthly by IV infusion over approximately 30 minutes. Participants in the present study received an OL weight-tiered dose of abatacept 10 mg/kg.
Arm/Group | OL Abatacept: Original 10 mg/kg | OL Abatacept: Original 2 mg/kg | OL Abatacept: Original Placebo
Number analyzed (Participants) | 84 | 68 | 67
mg/dL
  Baseline for Day 360 cohort (n=78, 65, 65) | 2.90 (2.25) | 3.02 (2.36) | 2.61 (2.20)
  Baseline for Day 720 cohort (n=68, 54, 53) | 2.64 (2.03) | 3.16 (2.60) | 2.60 (2.03)
  Baseline for Day 1080 cohort (n=61, 50, 47) | 2.58 (1.99) | 3.06 (2.63) | 2.52 (2.06)
  Baseline for Day 1440 cohort (n=56, 46, 41) | 2.65 (2.02) | 3.11 (2.71) | 2.62 (2.16)
  Baseline for Day 1800 cohort (n=52, 41, 41) | 2.40 (1.73) | 3.10 (2.75) | 2.64 (2.15)
  Baseline for Day 2160 cohort (n=43, 34, 33) | 2.34 (1.66) | 2.91 (2.77) | 2.80 (2.36)
  Baseline for Day 2520 cohort (n=36, 35, 32) | 2.46 (1.70) | 3.02 (2.79) | 2.86 (2.35)
  Baseline for Day 2880 cohort (n=27, 26, 27) | 2.14 (1.42) | 2.95 (3.00) | 3.08 (2.49)
  Baseline for Day 3060 cohort (n=14, 10, 8) | 1.93 (1.12) | 2.99 (3.07) | 2.72 (1.30)

48. Secondary Outcome: Mean Change From Baseline in Level of C Reactive Protein Over Time in OL Period
Description: Serum evaluations were carried out to evaluate participant concentrations of serum C reactive protein. Mean change from baseline=value at post-baseline OL time point-value and baseline OL time point.
Time Frame: Baseline (Day 0) and Days 360, 720, 1080, 1440, 1800, 2160, 2520, 2880, 3060
Population: as for outcome 18
Measure: Mean (Standard Error); unit: mg/dL
Groups:
- OL Abatacept: Original 2 mg/kg: Participants in the DB period received a weight-tiered dose of 2 mg/kg of abatacept that was administered monthly by an IV infusion over approximately 30 minutes. Participants in the present study received an OL weight-tiered dose of abatacept 10 mg/kg.
Arm/Group | OL Abatacept: Original 10 mg/kg | OL Abatacept: Original 2 mg/kg | OL Abatacept: Original Placebo
Number analyzed (Participants) | 84 | 68 | 67
mg/dL
  Change at Day 360 (n=78, 65, 65) | -1.38 (0.29) | -1.13 (0.33) | -0.08 (0.38)
  Change at Day 720 (n=68, 54, 53) | -1.46 (0.25) | -2.08 (0.38) | -1.26 (0.28)
  Change at Day 1080 (n=61, 50, 47) | -0.96 (0.44) | -1.93 (0.38) | -1.20 (0.35)
  Change at Day 1440 (n=56, 46, 41) | -1.56 (0.33) | -1.91 (0.37) | -1.21 (0.44)
  Change at Day 1800 (n=52, 41, 41) | -1.53 (0.25) | -1.33 (0.83) | -1.72 (0.35)
  Change at Day 2160 (n=43, 34, 33) | -1.33 (0.37) | -2.11 (0.46) | -2.04 (0.42)
  Change at Day 2520 (n=36, 35, 32) | -1.45 (0.39) | -2.29 (0.48) | -2.01 (0.40)
  Change at Day 2880 (n=27, 26, 27) | -1.47 (0.34) | -2.16 (0.61) | -2.25 (0.49)
  Change at Day 3060 (n=14, 10, 8) | -1.06 (0.36) | -2.10 (1.00) | -1.73 (0.50)

49. Secondary Outcome: Mean Baseline Physical Component Summary (PCS) of the Short-Form 36 (SF-36) Over Time in OL Period
Description: SF-36 = PCS & MCS & 8 individual indices (physical function, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, & mental health). Subscales were scored using norm-based methods that standardized scores to a mean of 50 & a standard deviation of 10 in the general population. Scores range from 0 to 100, with a higher score indicating better quality of life. Time-matched BL & post-BL values are presented for each post-BL visit & represent only that cohort with measurements available at that assessment. Change from BL data are presented in Outcome Measure 50.
Time Frame: Baseline (Day 0) and Days 360, 720, 1080, 1440, 1800, 2160, 2880, and 3060
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | OL Abatacept: Original 10 mg/kg | OL Abatacept: Original 2 mg/kg | OL Abatacept: Original Placebo
Number analyzed (Participants) | 84 | 68 | 67
Units on a Scale
  Baseline for Day 360 cohort (n=84, 66, 64) | 30.90 (8.14) | 31.03 (8.87) | 32.57 (7.94)
  Baseline for Day 720 cohort (n=73, 55, 53) | 31.44 (8.35) | 30.83 (8.03) | 32.48 (7.14)
  Baseline for Day 1080 cohort (n=63, 50, 49) | 31.56 (8.14) | 31.73 (8.63) | 32.38 (7.08)
  Baseline for Day 1440 cohort (n=59, 46, 44) | 31.46 (8.31) | 31.80 (8.84) | 32.20 (7.44)
  Baseline for Day 1800 cohort (n=54, 43, 42) | 32.19 (8.72) | 32.02 (8.91) | 32.36 (7.57)
  Baseline for Day 2160 cohort (n=45, 36, 35) | 32.15 (8.72) | 32.25 (9.07) | 32.29 (7.70)
  Baseline for Day 2520 cohort (n=38, 35, 33) | 31.93 (9.50) | 32.75 (9.20) | 32.54 (7.39)
  Baseline for Day 2880 cohort (n=33, 30, 31) | 32.63 (8.71) | 33.65 (8.66) | 32.66 (7.81)
  Baseline for Day 3060 cohort (n=17, 17, 16) | 36.81 (7.68) | 33.88 (9.12) | 33.40 (9.52)

50. Secondary Outcome: Mean Change From Baseline (BL) in the Physical Component Summary (PCS) of the SF-36 Over Time in OL Period
Description: The SF-36 consists of 2 summaries, the PCS and the MCS, and 8 individual indexes. The MCS addresses 4 of the 8 individual indices: vitality, social functioning, role-emotional, and mental health. The scores range from 0 to 100, with a higher score indicating better quality of life. Mean change from baseline=value at post-baseline OL time point-value and baseline OL time point. Baseline data for these time-matched cohorts are presented in Outcome Measure 49.
Time Frame: Baseline (Day 0) and Days 360, 720, 1080, 1440, 1800, 2160, 2880, and 3060
Population: as for outcome 38
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | OL Abatacept: Original 10 mg/kg | OL Abatacept: Original 2 mg/kg | OL Abatacept: Original Placebo
Number analyzed (Participants) | 84 | 68 | 67
Units on a Scale
  Change from BL on Day 360 (n=84, 66, 64) | 9.66 (1.05) | 7.13 (0.99) | 4.53 (1.04)
  Change from BL on Day 720 (n=73, 55, 53) | 9.15 (1.17) | 8.48 (1.25) | 8.30 (1.10)
  Change from BL on Day 1080 (n=63, 50, 49) | 9.28 (1.22) | 8.14 (1.36) | 9.28 (1.29)
  Change from BL on Day 1440 (n=59, 46, 44) | 8.18 (1.33) | 9.53 (1.28) | 9.50 (1.29)
  Change from BL on Day 1800 (n=54, 43, 42) | 9.30 (1.49) | 7.60 (1.25) | 9.18 (1.20)
  Change from BL on Day 2160 (n=45, 36, 35) | 9.51 (1.72) | 10.61 (1.44) | 8.86 (1.65)
  Change from BL on Day 2520 (n=38, 35, 33) | 10.12 (1.88) | 8.26 (1.58) | 7.92 (1.80)
  Change from BL on Day 2880 (n=33, 30, 31) | 10.97 (1.96) | 7.51 (1.35) | 9.19 (1.64)
  Change from BL on Day 3060 (n=17, 17, 16) | 8.55 (2.74) | 5.70 (1.98) | 9.06 (2.35)

51. Secondary Outcome: Mean Baseline Mental Component Summary (MCS) of the SF-36 Over Time in OL Period
Description: SF-36=PCS, MCS, & 8 individual indices. MCS addresses 4 of the 8 indices: vitality, social functioning, role-emotional, & mental health. Subscales were scored using norm-based methods that standardized the scores to a mean of 50 & a standard deviation of 10 in the general population. Scores range from 0 to 100, with a higher score indicating better quality of life. Time-matched baseline (Day 0) values & post-baseline (BL) values are presented for each post-BL visit & represent only that cohort with measurements available at that post-BL assessment. See Outcome Measure 51 for Change from BL.
Time Frame: Baseline (Day 0) and Days 360, 720, 1080, 1440, 1800, 2160, 2880, and 3060
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- OL Abatacept: Original Placebo: Participants in the double-blind period received a placebo administered monthly by IV infusion over approximately 30 minutes. Participants in the present study received an OL weight-tiered dose of abatacept 10 mg/kg.
Arm/Group | OL Abatacept: Original 10 mg/kg | OL Abatacept: Original 2 mg/kg | OL Abatacept: Original Placebo
Number analyzed (Participants) | 84 | 68 | 67
Units on a Scale
  Baseline (Day 0) for Day 360 cohort (n=84, 66, 64) | 46.27 (12.13) | 42.10 (13.08) | 44.44 (12.36)
  Baseline (Day 0) for Day 720 cohort (n=73,55, 53) | 46.17 (12.24) | 41.82 (13.10) | 44.74 (12.62)
  Baseline for Day 1080 cohort (n=63, 50, 49) | 45.45 (11.76) | 42.10 (12.82) | 44.53 (12.52)
  Baseline for Day 1440 cohort (n=59, 46, 44) | 45.32 (11.38) | 42.48 (13.06) | 44.66 (12.74)
  Baseline for Day 1800 cohort (n=54, 43, 42) | 45.07 (11.31) | 41.87 (12.99) | 44.68 (12.85)
  Baseline for Day 2160 cohort (n=45, 36, 35) | 45.57 (11.45) | 42.09 (12.96) | 43.89 (12.36)
  Baseline for Day 2520 cohort (n=38, 35, 33) | 46.35 (12.07) | 42.53 (13.34) | 44.51 (12.09)
  Baseline for Day 2880 cohort (n=33, 30, 31) | 45.48 (11.45) | 40.74 (12.02) | 43.51 (11.20)
  Baseline for Day 3060 cohort (n=17, 17, 16) | 46.24 (13.26) | 40.94 (13.47) | 45.14 (12.42)

52. Secondary Outcome: Mean Change From Baseline (BL) in the MCS of the SF-36 Over Time in OL Period
Description: The SF-36 consists of 2 summaries, the PCS and the MCS, and 8 individual indexes. The MCS addresses 4 of the 8 individual indices: vitality, social functioning, role-emotional, and mental health. The scores range from 0 to 100, with a higher score indicating better quality of life. Mean change from baseline=value at post-baseline OL time point-value and baseline OL time point. Baseline data for these time-matched cohorts are presented in Outcome Measure 51.
Time Frame: Baseline (Day 0) and Days 360, 450, 540, 630, 720, 810, 900, 1080, 1350, 1440, 1530, 1620, 1710, 1800, 1980, 2160, 2340, 2520, 2700, 2880, and 3060
Population: as for outcome 38
Measure: Mean (Standard Error); unit: Units on a Scale
Groups:
- OL Abatacept: Original 2 mg / kg Group: Participants in the DB period received a weight-tiered dose of 2 mg/kg of abatacept administered monthly by IV infusion over approximately 30 minutes. Participants in the present study received an OL weight-tiered dose of abatacept 10 mg/kg.
Arm/Group | OL Abatacept: Original 10 mg/kg | OL Abatacept: Original 2 mg / kg Group | OL Abatacept: Original Placebo
Number analyzed (Participants) | 84 | 68 | 67
Units on a Scale
  Change from BL at Day 360 (n=84, 66, 64) | 6.05 (1.19) | 6.03 (1.32) | 2.53 (1.34)
  Change from BL at Day 720 (n=73,55, 53) | 4.59 (1.29) | 6.02 (1.49) | 4.17 (1.57)
  Change from BL at Day 1080 (n=63, 50, 49) | 4.01 (1.23) | 4.87 (1.44) | 5.52 (1.78)
  Change from BL at Day 1440 (n=59, 46, 44) | 4.67 (1.31) | 6.68 (1.34) | 4.76 (2.12)
  Change from BL at Day 1800 (n=54, 43, 42) | 5.32 (1.38) | 4.59 (1.66) | 2.26 (1.71)
  Change from BL at Day 2160 (n=45, 36, 35) | 6.22 (1.47) | 5.95 (1.46) | 4.55 (2.19)
  Change from BL at Day 2520 (n=38, 35, 33) | 2.81 (1.85) | 7.34 (1.75) | 4.44 (2.26)
  Change from BL at Day 2880 (n=33, 30, 31) | 5.00 (1.92) | 6.97 (1.69) | 3.87 (2.18)
  Change from BL at Day 3060 (n=17, 17, 16) | 4.81 (2.90) | 5.51 (2.88) | 1.91 (3.26)

53. Secondary Outcome: Mean Baseline (BL) Physical Functioning Domain of the SF-36 Over Time in OL Period
Description: SF-36 = PCS & MCS & 8 individual indices (physical function, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, & mental health). Subscales were scored using norm-based methods that standardized scores to a mean of 50 & a standard deviation of 10 in the general population. Scores range from 0 to 100, with a higher score indicating better quality of life. Time-matched BL & post-BL values are presented for each post-BL visit & represent only that cohort with measurements available at that assessment. Change from BL data are presented in Outcome Measure 54.
Time Frame: Baseline (Day 0) and Days 360, 720, 1080, 1440, 1800, 2160, 2520, 2880, and 3060
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | OL Abatacept: Original 10 mg/kg | OL Abatacept: Original 2 mg/kg | OL Abatacept: Original Placebo
Number analyzed (Participants) | 84 | 68 | 67
Units on a Scale
  Baseline for Day 360 cohort (n=84, 67, 66) | 29.84 (9.57) | 30.18 (10.23) | 30.80 (9.48)
  Baseline for Day 720 cohort (n=73, 56, 53) | 30.39 (9.63) | 30.58 (9.99) | 30.79 (9.10)
  Baseline for Day 1080 cohort (n=64, 50, 49) | 30.27 (9.38) | 31.21 (10.35) | 30.95 (8.95)
  Baseline for Day 1440 cohort (n=60, 46, 44) | 30.47 (9.43) | 31.50 (10.12) | 31.26 (9.15)
  Baseline for Day 1800 cohort (n=54, 43, 42) | 30.96 (9.74) | 31.81 (10.45) | 31.48 (9.08)
  Baseline for Day 2160 cohort (n=45, 37, 35) | 31.41 (10.16) | 32.24 (10.42) | 31.56 (9.51)
  Baseline for Day 2520 cohort (n=38, 35, 33) | 31.47 (10.64) | 32.79 (10.26) | 32.04 (8.95)
  Baseline for Day 2880 cohort (n=33, 30, 31) | 31.77 (10.62) | 33.56 (10.07) | 32.18 (9.32)
  Baseline for Day 3060 cohort (n=18, 18, 16) | 34.97 (9.74) | 33.92 (9.55) | 32.37 (10.37)

54. Secondary Outcome: Mean Change From Baseline (BL) in the Physical Functioning Domain of the SF-36 Over Time in OL Period
Description: SF-36=2 summaries (PCS & MCS) & 8 individual indices including physical function, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, & mental health. All subscales were scored using norm-based methods that standardized the scores to a mean of 50 & a standard deviation of 10 in the general population. The scores range from 0 to 100, with a higher score indicating better quality of life. Mean change from BL = value at post-BL OL time point-value and BL OL time point. Baseline data for these time-matched cohorts are presented in Outcome Measure 53.
Time Frame: Baseline (Day 0) and Days 360, 720, 1080, 1440, 1800, 2160, 2520, 2880, and 3060
Population: as for outcome 38
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | OL Abatacept: Original 10 mg/kg | OL Abatacept: Original 2 mg/kg | OL Abatacept: Original Placebo
Number analyzed (Participants) | 84 | 68 | 67
Units on a Scale
  Change from BL at Day 360 (n=84, 67, 66) | 8.58 (1.11) | 6.53 (0.99) | 3.31 (0.92)
  Change from BL at Day 720 (n=73, 56, 53) | 8.36 (1.16) | 7.50 (1.32) | 7.30 (1.15)
  Change from BL at Day 1080 (n=64, 50, 49) | 8.36 (1.32) | 6.22 (1.49) | 7.62 (1.08)
  Change from BL at Day 1440 (n=60, 46, 44) | 7.91 (1.48) | 7.19 (1.48) | 7.58 (1.22)
  Change from BL at Day 1800 (n=54, 43, 42) | 8.39 (1.60) | 5.48 (1.45) | 6.16 (1.33)
  Change from BL at Day 2160 (n=45, 37, 35) | 9.24 (1.74) | 8.28 (1.53) | 5.46 (1.32)
  Change from BL at Day 2520 (n=38, 35, 33) | 7.92 (2.02) | 6.58 (1.74) | 5.87 (1.64)
  Change from BL at Day 2880 (n=33, 30, 31) | 9.93 (2.09) | 5.90 (1.63) | 6.63 (1.49)
  Change from BL at Day 3060 (n=18, 18, 16) | 6.21 (2.87) | 4.29 (1.91) | 6.16 (2.01)

55. Secondary Outcome: Mean Baseline Role-Physical Domain of the SF-36 Over Time in OL Period
Description: SF-36 = PCS & MCS & 8 individual indices (physical function, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, & mental health). Subscales were scored using norm-based methods that standardized scores to a mean of 50 & a standard deviation of 10 in the general population. Scores range from 0 to 100, with a higher score indicating better quality of life. Time-matched BL & post-BL values are presented for each post-BL visit & represent only that cohort with measurements available at that assessment. Change from BL data are presented in Outcome Measure 56.
Time Frame: Baseline (Day 0) and Days 360, 720, 1080, 1440, 1800, 2160, 2520, 2880, and 3060
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | OL Abatacept: Original 10 mg/kg | OL Abatacept: Original 2 mg/kg | OL Abatacept: Original Placebo
Number analyzed (Participants) | 84 | 68 | 67
Units on a Scale
  Baseline for Day 360 cohort (n=84, 66, 66) | 33.68 (9.66) | 31.70 (7.77) | 34.17 (8.82)
  Baseline for Day 720 cohort (n=73, 56, 53) | 34.06 (10.09) | 31.49 (7.51) | 33.69 (8.78)
  Baseline for Day 1080 cohort (n=64, 50, 49) | 34.36 (10.22) | 32.20 (7.96) | 33.58 (8.42)
  Baseline for Day 1440 cohort (n=60, 46, 44) | 33.97 (9.90) | 32.57 (8.20) | 33.10 (7.98)
  Baseline for Day 1800 cohort (n=54, 43, 42) | 33.85 (9.79) | 32.39 (8.31) | 33.01 (8.01)
  Baseline for Day 2160 cohort (n=45, 36, 35) | 33.61 (9.61) | 33.26 (8.85) | 32.80 (7.63)
  Baseline for Day 2520 cohort (n=38, 35, 33) | 33.72 (9.85) | 33.41 (8.93) | 33.95 (8.68)
  Baseline for Day 2880 cohort (n=33, 30, 31) | 33.74 (9.60) | 33.38 (8.45) | 33.43 (7.90)
  Baseline for Day 3060 cohort (n=17, 18, 16) | 37.52 (11.71) | 34.63 (8.57) | 35.47 (9.82)

56. Secondary Outcome: Mean Change From Baseline (BL) in the Role-Physical Domain of the SF-36 Over Time in OL Period
Description: SF-36=2 summaries (PCS & MCS) & 8 individual indices including physical function, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, & mental health. All subscales were scored using norm-based methods that standardized the scores to a mean of 50 & a standard deviation of 10 in the general population. The scores range from 0 to 100, with a higher score indicating better quality of life. Mean change from BL = value at post-BL OL time point-value and BL OL time point. Baseline data for these time-matched cohorts are presented in Outcome Measure 55.
Time Frame: Baseline (Day 0) and Days 360, 720, 1080, 1440, 1800, 2160, 2520, 2880, and 3060
Population: as for outcome 38
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | OL Abatacept: Original 10 mg/kg | OL Abatacept: Original 2 mg/kg | OL Abatacept: Original Placebo
Number analyzed (Participants) | 84 | 68 | 67
Units on a Scale
  Change from BL at Day 360 (n=84, 66, 66) | 10.10 (1.32) | 6.97 (1.22) | 5.68 (1.51)
  Change from BL at Day 720 (n=73, 56, 53) | 9.69 (1.51) | 9.60 (1.49) | 9.03 (1.55)
  Change from BL at Day 1080 (n=64, 50, 49) | 8.73 (1.63) | 8.06 (1.69) | 12.12 (1.86)
  Change from BL at Day 1440 (n=60, 46, 44) | 7.78 (1.69) | 10.30 (1.66) | 11.89 (1.76)
  Change from BL at Day 1800 (n=54, 43, 42) | 9.95 (1.85) | 7.57 (1.50) | 11.11 (1.74)
  Change from BL at Day 2160 (n=45, 36, 35) | 10.37 (1.86) | 10.41 (1.92) | 11.65 (2.14)
  Change from BL at Day 2520 (n=38, 35, 33) | 9.49 (2.20) | 9.50 (1.94) | 9.43 (2.57)
  Change from BL at Day 2880 (n=33, 30, 31) | 11.79 (2.32) | 7.31 (1.84) | 10.95 (2.32)
  Change from BL at Day 3060 (n=17, 18, 16) | 11.65 (3.53) | 4.32 (2.63) | 10.61 (3.48)

57. Secondary Outcome: Mean Baseline Bodily Pain Domain of the SF-36 Over Time in OL Period
Description: SF-36 = PCS & MCS & 8 individual indices (physical function, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, & mental health). Subscales were scored using norm-based methods that standardized scores to a mean of 50 & a standard deviation of 10 in the general population. Scores range from 0 to 100, with a higher score indicating better quality of life. Time-matched BL & post-BL values are presented for each post-BL visit & represent only that cohort with measurements available at that assessment. Change from BL data are presented in Outcome Measure 58.
Time Frame: Baseline (Day 0) and Days 360, 720, 1080, 1440, 1800, 2160, 2520, 2880, and 3060
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | OL Abatacept: Original 10 mg/kg | OL Abatacept: Original 2 mg/kg | OL Abatacept: Original Placebo
Number analyzed (Participants) | 84 | 68 | 67
Units on a Scale
  Baseline for Day 360 cohort (n=84, 67, 66) | 35.91 (8.52) | 33.82 (7.69) | 36.39 (7.98)
  Baseline for Day 720 cohort (n=73, 56, 53) | 36.10 (8.76) | 34.23 (7.63) | 35.93 (7.35)
  Baselinefor Day 1080 cohort (n=64, 50, 49) | 36.06 (8.73) | 34.57 (7.84) | 36.04 (7.48)
  Baseline for Day 1440 cohort (n=60, 46, 44) | 35.28 (8.59) | 34.56 (7.99) | 35.42 (7.37)
  Baseline for Day 1800 cohort (n=54, 43, 42) | 36.22 (8.94) | 34.57 (8.23) | 35.54 (7.27)
  Baseline for Day 2160 cohort (n=45, 36, 35) | 35.57 (9.35) | 34.50 (8.27) | 35.59 (7.65)
  Baseline for Day 2520 cohort (n=38, 35, 33) | 35.35 (9.49) | 35.29 (8.32) | 35.32 (7.73)
  Baseline for Day 2880 cohort (n=33, 30, 31) | 35.12 (9.68) | 35.76 (8.27) | 35.29 (8.03)
  Baseline for Day 3060 cohort (n=17, 18, 16) | 38.83 (9.60) | 35.75 (7.82) | 37.72 (8.69)

58. Secondary Outcome: Mean Change From BL in the Bodily Pain Domain of the SF-36 Over Time in OL Period
Description: SF-36=2 summaries (PCS & MCS) & 8 individual indices including physical function, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, & mental health. All subscales were scored using norm-based methods that standardized the scores to a mean of 50 & a standard deviation of 10 in the general population. The scores range from 0 to 100, with a higher score indicating better quality of life. Mean change from BL = value at post-BL OL time point-value and BL OL time point. Baseline data for these time-matched cohorts are presented in Outcome Measure 57.
Time Frame: BL (Day 0); Day 360; Day 720; Day 1,080; Day 1,440; Day 1,800; Day 2,160; Day 2,520; Day 2,880; Day 3,060
Population: as for outcome 40
Measure: Mean (Standard Error); unit: Units on a Scale
Groups:
- OL Abatacept: Original 10 mg / kg Group: Participants in the double-blind period received a weight-tiered dose of 10 mg/kg of abatacept that was administered monthly by an intravenous (IV) infusion over approximately 30 minutes. Participants weighing < 60 kg received abatacept 500 mg, participants weighing ≥ 60 kg and ≤ 100 kg received abatacept 750 mg, and participants > 100 kg received abatacept 1 g. Participants in the present study received an open-label weight-tiered dose of abatacept 10 mg/kg.
- OL Abatacept: Original 2 mg / kg Group: Participants in the double-blind period received a weight-tiered dose of 2 mg/kg of abatacept that was administered monthly by an intravenous (IV) infusion over approximately 30 minutes. Participants in the present study received an open-label weight-tiered dose of abatacept 10 mg/kg.
Arm/Group | OL Abatacept: Original 10 mg / kg Group | OL Abatacept: Original 2 mg / kg Group | OL Abatacept: Original Placebo Group
Number analyzed (Participants) | 84 | 68 | 67
Units on a Scale
  Change from BL at Day 360 (n=84, 67, 66) | 10.35 (1.14) | 9.26 (1.07) | 4.12 (1.13)
  Change from BL at Day 720 (n=73, 56, 53) | 8.84 (1.36) | 9.40 (1.33) | 9.17 (1.42)
  Change from BL at Day 1,080 (n=64, 50, 49) | 9.02 (1.35) | 9.67 (1.55) | 9.48 (1.59)
  Change from BL at Day 1,440 (n=60, 46, 44) | 9.54 (1.37) | 11.38 (1.59) | 10.86 (1.61)
  Change from BL at Day 1,800 (n=54, 43, 42) | 9.08 (1.50) | 8.73 (1.62) | 10.03 (1.64)
  Change from BL at Day 2,160 (n=45, 36, 35) | 10.27 (1.83) | 12.11 (1.66) | 10.83 (1.74)
  Change from BL at Day 2,520 (n=38, 35, 33) | 10.97 (1.90) | 10.55 (1.61) | 10.11 (1.76)
  Change from BL at Day 2,880 (n=33, 30, 31) | 11.68 (1.99) | 10.08 (1.66) | 10.86 (1.86)
  Change from BL at Day 3,060 (n=17, 18, 16) | 9.28 (3.77) | 6.45 (2.85) | 10.52 (3.15)

59. Secondary Outcome: Mean BL General Health Domain of the SF-36 Over Time in OL Period
Description: SF-36 = PCS & MCS & 8 individual indices (physical function, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, & mental health). Subscales were scored using norm-based methods that standardized scores to a mean of 50 & a standard deviation of 10 in the general population. Scores range from 0 to 100, with a higher score indicating better quality of life. Time-matched BL & post-BL values are presented for each post-BL visit & represent only that cohort with measurements available at that assessment. Change from BL data are presented in Outcome Measure 60.
Time Frame: Baseline (Day 0) and Days 360, 720, 1080, 1440, 1800, 2160, 2520, 2880, and 3060
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | OL Abatacept: Original 10 mg / kg Group | OL Abatacept: Original 2 mg / kg Group | OL Abatacept: Original Placebo Group
Number analyzed (Participants) | 84 | 68 | 67
Units on a Scale
  BL (Day 0) for Day 360 cohort (n=84, 67, 66) | 37.11 (9.23) | 35.87 (9.23) | 37.45 (9.01)
  BL (Day 0) for Day 720 cohort (n=73, 56, 53) | 37.36 (9.30) | 35.61 (8.96) | 38.06 (8.26)
  BL (Day 0) for Day 1,080 cohort (n=64, 50, 49) | 37.55 (9.38) | 35.78 (9.13) | 37.45 (8.37)
  BL (Day 0) for Day 1,440 cohort (n=60, 46, 44) | 37.41 (9.12) | 35.67 (8.88) | 37.64 (8.60)
  BL (Day 0) for Day 1,800 cohort (n=54, 43, 42) | 38.08 (9.75) | 35.60 (8.98) | 37.78 (8.59)
  BL (Day 0) for Day 2,160 cohort (n=45, 37, 35) | 38.81 (9.94) | 35.69 (8.85) | 36.93 (8.65)
  BL (Day 0) for Day 2,520 cohort (n=38, 36, 33) | 39.25 (10.40) | 36.17 (9.40) | 36.98 (8.50)
  BL (Day 0) for Day 2,880 cohort (n=33, 30, 31) | 40.09 (10.49) | 35.39 (8.54) | 36.57 (8.54)
  BL (Day 0) for Day 3,060 cohort (n=18, 18, 16) | 41.37 (11.49) | 33.88 (8.58) | 36.84 (9.18)

60. Secondary Outcome: Mean Change From Baseline (BL) in the General Health Domain of the SF-36 Over Time in OL Period
Description: SF-36=2 summaries (PCS & MCS) & 8 individual indices including physical function, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, & mental health. All subscales were scored using norm-based methods that standardized the scores to a mean of 50 & a standard deviation of 10 in the general population. The scores range from 0 to 100, with a higher score indicating better quality of life. Mean change from BL = value at post-BL OL time point-value and BL OL time point. Baseline data for these time-matched cohorts are presented in Outcome Measure 59.
Time Frame: Baseline (Day 0) and Days 360, 720, 1080, 1440, 1800, 2160, 2520, 2880, and 3060
Population: as for outcome 18
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | OL Abatacept: Original 10 mg/kg | OL Abatacept: Original 2 mg/kg | OL Abatacept: Original Placebo
Number analyzed (Participants) | 84 | 68 | 67
Units on a Scale
  Change from BL at Day 360 (n=84, 67, 66) | 6.98 (0.90) | 6.08 (1.05) | 3.48 (0.71)
  Change from BL at Day 720 (n=73, 56, 53) | 5.96 (1.06) | 5.99 (1.24) | 5.09 (0.96)
  Change from BL at Day 1080 (n=64, 50, 49) | 6.18 (1.12) | 6.27 (1.07) | 5.63 (1.05)
  Change from BL at Day 1440 (n=60, 46, 44) | 5.84 (1.12) | 8.01 (0.91) | 4.80 (1.17)
  Change from BL at Day 1800 (n=54, 43, 42) | 6.52 (1.25) | 6.87 (1.26) | 3.97 (1.25)
  Change from BL at Day 2160 (n=45, 37, 35) | 5.27 (1.40) | 8.73 (1.30) | 5.38 (1.56)
  Change from BL at Day 2520 (n=38, 36, 33) | 6.42 (1.85) | 6.51 (1.21) | 5.38 (1.43)
  Change from BL at Day 2880 (n=33, 30, 31) | 6.37 (2.05) | 8.67 (1.45) | 5.61 (1.30)
  Change from BL at Day 3060 (n=18, 18, 16) | 5.09 (2.73) | 6.82 (2.21) | 3.88 (1.46)

61. Secondary Outcome: Mean Baseline Vitality Domain of the SF-36 Over Time in OL Period
Description: SF-36 = PCS & MCS & 8 individual indices (physical function, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, & mental health). Subscales were scored using norm-based methods that standardized scores to a mean of 50 & a standard deviation of 10 in the general population. Scores range from 0 to 100, with a higher score indicating better quality of life. Time-matched BL & post-BL values are presented for each post-BL visit & represent only that cohort with measurements available at that assessment. Change from BL data are presented in Outcome Measure 62.
Time Frame: Baseline (Day 0) and Days 360, 720, 1080, 1440, 1800, 2160, 2520, 2880, and 3060
Population: All treated OL participants. Participants were grouped according to the treatment they received in the DB study. n = the number of participants with measurements for that time point.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- OL Abatacept: Original 10 mg/kg: Participants in the DB period received a weight-tiered dose of 10 mg/kg of abatacept administered monthly by an IV infusion over approximately 30 minutes. Participants weighing <60 kg received abatacept 500 mg, participants weighing ≥60 kg and ≤100 kg received abatacept 750 mg, and participants >100 kg received abatacept 1 g. Participants in the present study received an OL weight-tiered dose of abatacept 10 mg/kg.
- OL Abatacept: Original 2 mg/kg: Participants in the DB period received a weight-tiered dose of 2 mg/kg of abatacept that was administered monthly by IV infusion over approximately 30 minutes. Participants in the present study received an open-label weight-tiered dose of abatacept 10 mg/kg.
- OL Abatacept: Original Placebo: Participants in the double-blind period received a placebo that was administered monthly by IV infusion over approximately 30 minutes. Participants in the present study received an OL weight-tiered dose of abatacept 10 mg/kg.
Arm/Group | OL Abatacept: Original 10 mg/kg | OL Abatacept: Original 2 mg/kg | OL Abatacept: Original Placebo
Number analyzed (Participants) | 84 | 68 | 67
Units on a Scale
  Baseline for Day 360 cohort (n=84, 67, 66) | 41.17 (8.29) | 40.68 (8.84) | 42.49 (9.81)
  Baseline for Day 720 cohort (n=73, 55, 53) | 41.15 (8.29) | 41.22 (8.25) | 43.25 (9.84)
  Baseline for Day 1080 cohort (n=63, 50, 49) | 40.65 (8.24) | 41.72 (8.56) | 42.58 (9.81)
  Baseline for Day 1440 cohort (n=59, 46, 44) | 40.84 (8.17) | 41.85 (8.81) | 43.08 (9.81)
  Baseline for Day 1800 cohort (n=54, 43, 42) | 41.09 (8.27) | 41.40 (8.72) | 43.42 (9.83)
  Baseline for Day 2160 cohort (n=45, 37, 35) | 41.66 (8.59) | 40.93 (8.65) | 42.77 (10.04)
  Baseline for Day 2520 cohort (n=38, 36, 33) | 41.66 (9.03) | 41.43 (9.26) | 42.74 (9.64)
  Baseline for Day 2880 cohort (n=33, 30, 31) | 42.12 (8.80) | 40.22 (8.22) | 42.34 (9.57)
  Baseline for Day 3060 cohort (n=18, 17, 16) | 44.06 (8.66) | 41.12 (7.29) | 42.40 (9.20)

62. Secondary Outcome: Mean Change From Baseline (BL) in the Vitality Domain of the SF-36 Over Time in OL Period
Description: SF-36=2 summaries (PCS & MCS) & 8 individual indices including physical function, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, & mental health. All subscales were scored using norm-based methods that standardized the scores to a mean of 50 & a standard deviation of 10 in the general population. The scores range from 0 to 100, with a higher score indicating better quality of life. Mean change from BL = value at post-BL OL time point-value and BL OL time point. Baseline data for these time-matched cohorts are presented in Outcome Measure 61.
Time Frame: Baseline (Day 0) and Days 360, 720, 1080, 1440, 1800, 2160, 2520, 2880, and 3060
Population: as for outcome 38
Measure: Mean (Standard Error); unit: Units on a Scale
Groups:
- OL Abatacept: Original 10 mg /kg: Participants in the DB period received a weight-tiered dose of 10 mg/kg of abatacept that was administered monthly by IV infusion over approximately 30 minutes. Participants weighing <60 kg received abatacept 500 mg, participants weighing ≥60 kg and ≤100 kg received abatacept 750 mg, and participants >100 kg received abatacept 1 g. Participants in the present study received an OL weight-tiered dose of abatacept 10 mg/kg.
Arm/Group | OL Abatacept: Original 10 mg /kg | OL Abatacept: Original 2 mg/kg | OL Abatacept: Original Placebo
Number analyzed (Participants) | 84 | 68 | 67
Units on a Scale
  Change from BL at Day 360 (n=84, 67, 66) | 8.50 (1.02) | 4.91 (1.03) | 1.86 (1.04)
  Change from BL at Day 720 (n=73, 55, 53) | 7.77 (1.01) | 6.20 (1.27) | 4.69 (1.20)
  Change from BL at Day 1080 (n=63, 50, 49) | 7.73 (1.18) | 6.30 (1.16) | 6.46 (1.23)
  Change from BL at Day 1440 (n=59, 46, 44) | 6.00 (1.25) | 7.61 (1.23) | 4.73 (1.62)
  Change from BL at Day 1800 (n=54, 43, 42) | 7.44 (1.41) | 6.33 (1.14) | 3.49 (1.70)
  Change from BL at Day 2160 (n=45, 37, 35) | 8.15 (1.53) | 7.10 (1.18) | 4.60 (1.96)
  Change from BL at Day 2520 (n=38, 36, 33) | 6.64 (1.98) | 6.86 (1.21) | 3.82 (2.03)
  Change from BL at Day 2880 (n=33, 30, 31) | 6.65 (1.86) | 7.10 (1.34) | 4.76 (1.70)
  Change from BL at Day 3060 (n=18, 17, 16) | 4.60 (3.02) | 6.68 (2.21) | 3.99 (2.34)

63. Secondary Outcome: Mean Baseline Social Functioning Domain of the SF-36 Over Time in OL Period
Description: SF-36 = PCS & MCS & 8 individual indices (physical function, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, & mental health). Subscales were scored using norm-based methods that standardized scores to a mean of 50 & a standard deviation of 10 in the general population. Scores range from 0 to 100, with a higher score indicating better quality of life. Time-matched BL & post-BL values are presented for each post-BL visit & represent only that cohort with measurements available at that assessment. Change from BL data are presented in Outcome Measure 64.
Time Frame: Baseline (Day 0) and Days 360, 720, 1080, 1440, 1800, 2160, 2520, 2880, and 3060
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- OL Abatacept: Original Placebo Group: Participants in the DB period received a placebo administered monthly by IV infusion over approximately 30 minutes. Participants in the present study received an OL weight-tiered dose of abatacept 10 mg/kg.
Arm/Group | OL Abatacept: Original 10 mg/kg | OL Abatacept: Original 2 mg/kg | OL Abatacept: Original Placebo Group
Number analyzed (Participants) | 84 | 68 | 67
Units on a Scale
  Baseline for Day 360 cohort (n=84, 67, 66) | 38.59 (10.99) | 34.45 (10.52) | 38.14 (10.91)
  Baseline for Day 720 cohort (n=73, 56, 53) | 39.37 (11.13) | 35.04 (9.81) | 39.11 (10.74)
  Baseline for Day 1080 cohort (n=64, 50, 49) | 38.99 (11.04) | 34.77 (9.22) | 39.08 (10.71)
  Baseline for Day 1440 cohort (n=60, 46, 44) | 38.77 (11.04) | 35.19 (9.36) | 38.88 (11.05)
  Baseline for Day 1800 cohort (n=54, 43, 42) | 38.84 (11.52) | 34.92 (9.54) | 39.04 (11.03)
  Baseline for Day 2160 cohort (n=45, 36, 35) | 39.16 (11.45) | 35.42 (9.54) | 38.06 (10.97)
  Baseline for Day 2520 cohort (n=38, 35, 33) | 39.42 (11.82) | 35.11 (9.85) | 38.88 (10.93)
  Baseline for Day 2880 cohort (n=33, 30, 31) | 39.54 (12.14) | 36.33 (8.80) | 38.40 (10.75)
  Baseline for Day 3060 cohort (n=17, 18, 16) | 42.77 (11.66) | 36.33 (8.78) | 38.82 (12.52)

64. Secondary Outcome: Mean Change From Baseline (BL) in the Social Functioning Domain of the SF-36 Over Time in OL Period
Description: SF-36=2 summaries (PCS & MCS) & 8 individual indices including physical function, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, & mental health. All subscales were scored using norm-based methods that standardized the scores to a mean of 50 & a standard deviation of 10 in the general population. The scores range from 0 to 100, with a higher score indicating better quality of life. Mean change from BL = value at post-BL OL time point-value and BL OL time point. Baseline data for these time-matched cohorts are presented in Outcome Measure 63.
Time Frame: Baseline (Day 0) and Days 360, 720, 1080, 1440, 1800, 2160, 2520, 2880, and 3060
Population: as for outcome 61
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | OL Abatacept: Original 10 mg/kg | OL Abatacept: Original 2 mg/kg | OL Abatacept: Original Placebo
Number analyzed (Participants) | 84 | 68 | 67
Units on a Scale
  Change from BL at Day 360 (n=84, 67, 66) | 8.47 (1.25) | 8.02 (1.11) | 4.44 (1.12)
  Change from BL at Day 720 (n=73, 56, 53) | 6.62 (1.39) | 8.43 (1.35) | 6.86 (1.28)
  Change from BL at Day 1080 (n=64, 50, 49) | 5.94 (1.20) | 8.25 (1.05) | 7.87 (1.38)
  Change from BL at Day 1440 (n=60, 46, 44) | 6.24 (1.51) | 9.56 (1.39) | 8.02 (1.82)
  Change from BL at Day 1800 (n=54, 43, 42) | 8.65 (1.49) | 6.69 (1.56) | 6.59 (1.86)
  Change from BL at Day 2160 (n=45, 36, 35) | 9.53 (1.58) | 9.95 (1.29) | 7.13 (2.08)
  Change from BL at Day 2520 (n=38, 35, 33) | 5.00 (2.24) | 10.70 (1.40) | 5.76 (2.19)
  Change from BL at Day 2880 (n=33, 30, 31) | 7.90 (1.99) | 6.69 (1.70) | 5.25 (1.93)
  Change from BL at Day 3060 (n=17, 18, 16) | 6.07 (2.98) | 6.03 (2.23) | 4.07 (3.03)

65. Secondary Outcome: Mean Baseline Role-Emotional Domain of the SF-36 Over Time in OL Period
Description: SF-36 = PCS & MCS & 8 individual indices (physical function, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, & mental health). Subscales were scored using norm-based methods that standardized scores to a mean of 50 & a standard deviation of 10 in the general population. Scores range from 0 to 100, with a higher score indicating better quality of life. Time-matched BL & post-BL values are presented for each post-BL visit & represent only that cohort with measurements available at that assessment. Change from BL data are presented in Outcome Measure 66.
Time Frame: Baseline (Day 0) and Days 360, 720, 1080, 1440, 1800, 2160, 2520, 2880, and 3060
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | OL Abatacept: Original 10 mg/kg | OL Abatacept: Original 2 mg/kg | OL Abatacept: Original Placebo
Number analyzed (Participants) | 84 | 68 | 67
Units on a Scale
  Baseline for Day 360 cohort (n=84, 67, 64) | 40.29 (14.09) | 36.63 (14.30) | 38.88 (14.28)
  Baseline for Day 720 cohort (n=73, 56, 53) | 40.19 (14.04) | 36.15 (14.08) | 38.84 (14.68)
  Baseline for Day 1080 cohort (n=64, 50, 49) | 39.21 (13.92) | 37.01 (14.09) | 39.43 (14.76)
  Baseline for Day 1440 cohort (n=60, 46, 44) | 38.84 (13.90) | 37.48 (14.02) | 39.30 (14.81)
  Baseline for Day 1800 cohort (n=54, 43, 42) | 38.76 (13.97) | 36.97 (14.19) | 39.29 (14.76)
  Baseline for Day 2160 cohort (n=45, 36, 35) | 38.72 (14.29) | 37.78 (14.02) | 39.09 (14.97)
  Baseline for Day 2520 cohort (n=38, 35, 33) | 39.54 (14.85) | 37.88 (14.21) | 40.34 (14.67)
  Baseline for Day 2880 cohort (n=33, 30, 31) | 38.10 (14.62) | 36.73 (14.29) | 39.37 (14.62)
  Baseline for Day 3060 cohort (n=17, 18, 16) | 40.47 (14.93) | 37.78 (14.45) | 44.15 (14.12)

66. Secondary Outcome: Mean Change From Baseline (BL) in the Role-Emotional Domain of the SF-36 Over Time in OL Period
Description: SF-36=2 summaries (PCS & MCS) & 8 individual indices including physical function, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, & mental health. All subscales were scored using norm-based methods that standardized the scores to a mean of 50 & a standard deviation of 10 in the general population. The scores range from 0 to 100, with a higher score indicating better quality of life. Mean change from BL = value at post-BL OL time point-value and BL OL time point. Baseline data for these time-matched cohorts are presented in Outcome Measure 65.
Time Frame: Baseline (Day 0) and Days 360, 720, 1080, 1440, 1800, 2160, 2520, 2880, and 3060
Population: as for outcome 61
Measure: Mean (Standard Error); unit: Units on a Scale
Groups:
- OL Abatacept: Original 10 mg/kg: Participants in the DB period received a weight-tiered dose of 10 mg/kg of abatacept that was administered monthly by an IV infusion over approximately 30 minutes. Participants weighing <60 kg received abatacept 500 mg, participants weighing ≥60 kg and ≤100 kg received abatacept 750 mg, and participants >100 kg received abatacept 1 g. Participants in the present study received an OL weight-tiered dose of abatacept 10 mg/kg.
- OL Abatacept: Original 2 mg/kg: Participants in the DBperiod received a weight-tiered dose of 2 mg/kg of abatacept administered monthly by IV infusion over approximately weight-tiered dose of abatacept 10 mg/kg.
Arm/Group | OL Abatacept: Original 10 mg/kg | OL Abatacept: Original 2 mg/kg | OL Abatacept: Original Placebo
Number analyzed (Participants) | 84 | 68 | 67
Units on a Scale
  Change from BL at Day 360 (n=84, 67, 64) | 8.03 (1.58) | 7.55 (2.05) | 3.79 (1.94)
  Change from BL at Day 720 (n=73, 56, 53) | 6.93 (1.68) | 8.28 (2.29) | 6.36 (1.97)
  Change from BL at Day 1080 (n=64, 50, 49) | 5.76 (1.88) | 4.64 (2.24) | 7.95 (2.27)
  Change from BL at Day 1440 (n=60, 46, 44) | 6.67 (1.86) | 8.24 (2.31) | 7.18 (2.56)
  Change from BL at Day 1800 (n=54, 43, 42) | 7.41 (2.04) | 4.16 (2.48) | 4.51 (2.19)
  Change from BL at Day 2160 (n=45, 36, 35) | 7.84 (2.16) | 7.61 (2.40) | 6.47 (2.87)
  Change from BL at Day 2520 (n=38, 35, 33) | 5.82 (2.34) | 8.43 (2.92) | 5.75 (2.64)
  Change from BL at Day 2880 (n=33, 30, 31) | 8.94 (2.72) | 8.78 (2.32) | 4.76 (3.04)
  Change from BL at Day 3060 (n=17, 18, 16) | 9.92 (4.09) | 5.85 (3.92) | 0.66 (4.66)

67. Secondary Outcome: Mean Baseline Mental Health Domain of the SF-36 Over Time in OL Period
Description: SF-36 = PCS & MCS & 8 individual indices (physical function, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, & mental health). Subscales were scored using norm-based methods that standardized scores to a mean of 50 & a standard deviation of 10 in the general population. Scores range from 0 to 100, with a higher score indicating better quality of life. Time-matched BL & post-BL values are presented for each post-BL visit & represent only that cohort with measurements available at that assessment. Change from BL data are presented in Outcome Measure 68.
Time Frame: Baseline (Day 0) and Days 360, 720, 1080, 1440, 1800, 2160, 2520, 2880, and 3060
Population: as for outcome 61
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | OL Abatacept: Original 10 mg/kg | OL Abatacept: Original 2 mg/kg | OL Abatacept: Original Placebo
Number analyzed (Participants) | 84 | 68 | 67
Units on a Scale
  Baseline for Day 360 cohort (n=84, 67, 66) | 44.66 (11.94) | 41.29 (12.28) | 42.35 (11.62)
  Baseline for Day 720 cohort (n=73, 55, 53) | 44.53 (12.19) | 40.49 (12.72) | 41.99 (11.58)
  Baseline for Day 1080 cohort (n=63, 50, 49) | 44.13 (11.82) | 40.81 (12.66) | 41.44 (11.55)
  Baseline for Day 1440 cohort (n=59, 46, 44) | 44.24 (11.09) | 41.11 (12.61) | 41.60 (11.77)
  Baseline for Day 1800 cohort (n=54, 43, 42) | 44.13 (11.14) | 40.78 (12.39) | 41.50 (11.78)
  Baseline for Day 2160 cohort (n=45, 37, 35) | 44.79 (11.18) | 40.50 (12.17) | 40.89 (11.05)
  Baselinefor Day 2520 cohort (n=38, 36, 33) | 45.54 (11.10) | 42.05 (12.54) | 41.06 (11.44)
  Baseline for Day 2880 cohort (n=33, 30, 31) | 44.87 (9.92) | 39.77 (10.76) | 40.24 (10.92)
  Baseline for Day 3060 cohort (n=18, 17, 16) | 44.89 (11.85) | 39.49 (11.62) | 40.18 (12.07)

68. Secondary Outcome: Mean Change From Baseline (BL) in the Mental Health Domain of the SF-36 Over Time in OL Period
Description: SF-36=2 summaries (PCS & MCS) & 8 individual indices including physical function, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, & mental health. All subscales were scored using norm-based methods that standardized the scores to a mean of 50 & a standard deviation of 10 in the general population. The scores range from 0 to 100, with a higher score indicating better quality of life. Mean change from BL = value at post-BL OL time point-value and BL OL time point. Baseline data for these time-matched cohorts are presented in Outcome Measure 67.
Time Frame: Baseline (Day 0) and Days 360, 720, 1080, 1440, 1800, 2160, 2520, 2880, and 3060
Population: as for outcome 40
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | OL Abatacept: Original 10 mg/kg | OL Abatacept: Original 2 mg/kg | OL Abatacept: Original Placebo
Number analyzed (Participants) | 84 | 68 | 67
Units on a Scale
  Change from BL at Day 360 (n=84, 67, 66) | 5.41 (1.10) | 5.74 (1.14) | 2.60 (1.13)
  Change from BL at Day 720 (n=73, 55, 53) | 4.22 (1.18) | 5.49 (1.29) | 4.59 (1.50)
  Change from BL at Day 1080 (n=63, 50, 49) | 4.62 (1.03) | 5.41 (1.48) | 5.54 (1.59)
  Change from BL at Day 1440 (n=59, 46, 44) | 4.81 (1.14) | 5.96 (1.24) | 5.59 (1.93)
  Change from BL at Day 1800 (n=54, 43, 42) | 4.47 (1.34) | 5.44 (1.45) | 3.15 (1.80)
  Change from BL at Day 2160 (n=45, 37, 35) | 5.82 (1.33) | 5.96 (1.26) | 5.29 (1.94)
  Change from BL at Day 2520 (n=38, 36, 33) | 3.15 (1.92) | 6.06 (1.50) | 6.33 (1.94)
  Change from BL at Day 2880 (n=33, 30, 31) | 4.96 (1.71) | 6.30 (1.60) | 6.78 (1.98)
  Change from BL at Day 3060 (n=18, 17, 16) | 2.65 (2.35) | 4.68 (2.59) | 6.99 (2.68)

ADVERSE EVENTS:
Arm/Group | Aba 10mg/kg+MTX | Aba 2mg/kg+MTX | Abatacept (LT) | Placebo+MTX
Serious Adverse Events (participants affected / at risk) | 17/115 | 19/105 | 117/219 | 21/119
Other Adverse Events (participants affected / at risk) | 96/115 | 98/105 | 200/219 | 108/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aba 10mg/kg+MTX (N=115) | Aba 2mg/kg+MTX (N=105) | Abatacept (LT) (N=219) | Placebo+MTX (N=119)
IRITIS (Eye disorders) | 0 | 0 | 1 | 0
ARTHROSCOPY (Investigations) | 0 | 1 | 0 | 0
SLEEP STUDY (Investigations) | 0 | 0 | 1 | 0
INVESTIGATION (Investigations) | 0 | 0 | 2 | 0
VASCULAR TEST (Investigations) | 0 | 0 | 1 | 0
ARTERIOGRAM CORONARY (Investigations) | 0 | 0 | 1 | 0
HAEMOGLOBIN DECREASED (Investigations) | 0 | 0 | 1 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 0 | 1 | 0
PERICARDITIS (Cardiac disorders) | 0 | 1 | 2 | 0
ANGINA PECTORIS (Cardiac disorders) | 0 | 0 | 1 | 1
ANGINA UNSTABLE (Cardiac disorders) | 1 | 0 | 1 | 0
CARDIAC ANEURYSM (Cardiac disorders) | 0 | 0 | 1 | 0
PLEUROPERICARDITIS (Cardiac disorders) | 0 | 0 | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 1 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 0 | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 3 | 1
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 | 0 | 1 | 0
CARDIOPULMONARY FAILURE (Cardiac disorders) | 0 | 0 | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 0 | 2 | 0
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 | 0 | 1 | 0
AORTIC VALVE INCOMPETENCE (Cardiac disorders) | 0 | 0 | 1 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 0 | 3 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0 | 1 | 0
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 0 | 1 | 1
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 0 | 0 | 1 | 0
EMBOLISM (Vascular disorders) | 0 | 0 | 1 | 0
HAEMATOMA (Vascular disorders) | 0 | 0 | 2 | 0
THROMBOSIS (Vascular disorders) | 0 | 0 | 1 | 0
HYPERTENSION (Vascular disorders) | 0 | 0 | 1 | 0
AORTIC ANEURYSM (Vascular disorders) | 1 | 0 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 4 | 0
AORTIC ANEURYSM RUPTURE (Vascular disorders) | 0 | 0 | 1 | 0
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 0 | 0 | 1 | 0
SUPERIOR VENA CAVAL OCCLUSION (Vascular disorders) | 0 | 0 | 1 | 0
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 | 0 | 1 | 0
JOINT PROSTHESIS USER (Social circumstances) | 1 | 0 | 0 | 0
ANXIETY (Psychiatric disorders) | 1 | 0 | 0 | 0
MAJOR DEPRESSION (Psychiatric disorders) | 0 | 0 | 1 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 0 | 1 | 0
BILIARY COLIC (Hepatobiliary disorders) | 0 | 0 | 2 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0 | 4 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 | 0 | 0 | 0
POLYARTERITIS NODOSA (Immune system disorders) | 0 | 0 | 1 | 0
SYNCOPE (Nervous system disorders) | 0 | 0 | 1 | 0
SCIATICA (Nervous system disorders) | 0 | 0 | 0 | 1
DIZZINESS (Nervous system disorders) | 0 | 1 | 1 | 0
CONVULSION (Nervous system disorders) | 0 | 0 | 1 | 0
HYPOAESTHESIA (Nervous system disorders) | 0 | 0 | 1 | 0
RADICULOPATHY (Nervous system disorders) | 0 | 0 | 1 | 0
RADICULAR PAIN (Nervous system disorders) | 0 | 0 | 1 | 0
PARTIAL SEIZURES (Nervous system disorders) | 0 | 0 | 1 | 0
MULTIPLE SCLEROSIS (Nervous system disorders) | 0 | 0 | 1 | 0
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 | 0 | 0 | 1
CEREBRAL ARTERY EMBOLISM (Nervous system disorders) | 0 | 0 | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 0 | 2 | 0
TRANSIENT GLOBAL AMNESIA (Nervous system disorders) | 0 | 0 | 1 | 0
CEREBELLAR ARTERY THROMBOSIS (Nervous system disorders) | 0 | 0 | 1 | 0
COLITIS (Gastrointestinal disorders) | 0 | 0 | 1 | 0
VOMITING (Gastrointestinal disorders) | 0 | 0 | 1 | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 1 | 1 | 0
GASTRIC ULCER (Gastrointestinal disorders) | 0 | 0 | 1 | 0
ABDOMINAL MASS (Gastrointestinal disorders) | 0 | 1 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 3 | 0
DUODENAL ULCER (Gastrointestinal disorders) | 0 | 0 | 1 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 1 | 1 | 0
UMBILICAL HERNIA (Gastrointestinal disorders) | 0 | 0 | 2 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 | 0 | 1 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1 | 0
HERNIAL EVENTRATION (Gastrointestinal disorders) | 0 | 0 | 1 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 0 | 1 | 0
OESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 0 | 0 | 1 | 0
PANCREATITIS CHRONIC (Gastrointestinal disorders) | 0 | 0 | 1 | 0
MALLORY-WEISS SYNDROME (Gastrointestinal disorders) | 0 | 0 | 1 | 0
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 1 | 0 | 0 | 0
RETROPERITONEAL HAEMATOMA (Gastrointestinal disorders) | 0 | 0 | 1 | 0
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0 | 0
UMBILICAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 0 | 0 | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
SEPSIS (Infections and infestations) | 0 | 0 | 0 | 1
ABSCESS (Infections and infestations) | 0 | 0 | 3 | 0
CYSTITIS (Infections and infestations) | 0 | 0 | 1 | 0
VIRAEMIA (Infections and infestations) | 0 | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 0 | 8 | 1
SINUSITIS (Infections and infestations) | 0 | 1 | 1 | 0
BRONCHITIS (Infections and infestations) | 1 | 0 | 0 | 0
CELLULITIS (Infections and infestations) | 0 | 1 | 1 | 0
ERYSIPELAS (Infections and infestations) | 0 | 0 | 2 | 0
OSTEOMYELITIS (Infections and infestations) | 0 | 1 | 0 | 0
DIVERTICULITIS (Infections and infestations) | 0 | 0 | 3 | 0
OTITIS EXTERNA (Infections and infestations) | 0 | 0 | 1 | 0
PYELONEPHRITIS (Infections and infestations) | 0 | 0 | 1 | 0
TOOTH INFECTION (Infections and infestations) | 0 | 0 | 1 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 0 | 0 | 1 | 0
AMOEBIC DYSENTERY (Infections and infestations) | 0 | 0 | 1 | 0
ESCHERICHIA SEPSIS (Infections and infestations) | 0 | 0 | 1 | 0
ARTHRITIS BACTERIAL (Infections and infestations) | 0 | 0 | 2 | 0
ARTHRITIS INFECTIVE (Infections and infestations) | 0 | 0 | 0 | 1
INFECTED SKIN ULCER (Infections and infestations) | 0 | 0 | 1 | 0
LOCALISED INFECTION (Infections and infestations) | 0 | 1 | 0 | 0
EYE INFECTION FUNGAL (Infections and infestations) | 0 | 0 | 1 | 0
PNEUMONIA HAEMOPHILUS (Infections and infestations) | 0 | 0 | 1 | 0
ABDOMINAL WALL ABSCESS (Infections and infestations) | 0 | 0 | 1 | 0
PERICARDITIS INFECTIVE (Infections and infestations) | 0 | 0 | 1 | 0
INTERVERTEBRAL DISCITIS (Infections and infestations) | 0 | 0 | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1 | 0
BACTERIAL PYELONEPHRITIS (Infections and infestations) | 0 | 0 | 1 | 0
DEVICE RELATED INFECTION (Infections and infestations) | 0 | 0 | 1 | 0
POST PROCEDURAL INFECTION (Infections and infestations) | 0 | 0 | 1 | 0
PROTEINURIA (Renal and urinary disorders) | 0 | 0 | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 0 | 0 | 1 | 0
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 | 0 | 1 | 0
ANGIOPLASTY (Surgical and medical procedures) | 0 | 1 | 0 | 0
ARTHRODESIS (Surgical and medical procedures) | 0 | 0 | 1 | 0
POLYPECTOMY (Surgical and medical procedures) | 1 | 0 | 0 | 0
SYNOVECTOMY (Surgical and medical procedures) | 0 | 1 | 0 | 1
CYST REMOVAL (Surgical and medical procedures) | 1 | 0 | 0 | 0
TENDON GRAFT (Surgical and medical procedures) | 0 | 0 | 0 | 1
STERILISATION (Surgical and medical procedures) | 0 | 0 | 1 | 0
FOOT OPERATION (Surgical and medical procedures) | 0 | 0 | 0 | 1
KNEE OPERATION (Surgical and medical procedures) | 0 | 0 | 1 | 0
BUNION OPERATION (Surgical and medical procedures) | 0 | 0 | 1 | 0
HIP ARTHROPLASTY (Surgical and medical procedures) | 1 | 0 | 3 | 0
KNEE ARTHROPLASTY (Surgical and medical procedures) | 0 | 1 | 0 | 1
JOINT ARTHROPLASTY (Surgical and medical procedures) | 0 | 1 | 0 | 0
CHOLESTEATOMA REMOVAL (Surgical and medical procedures) | 0 | 0 | 1 | 0
CORONARY ARTERY BYPASS (Surgical and medical procedures) | 0 | 1 | 0 | 0
MITRAL VALVE REPLACEMENT (Surgical and medical procedures) | 0 | 1 | 0 | 0
GOUT (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
DIABETIC FOOT (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
LYMPHOID TISSUE HYPERPLASIA (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
MENORRHAGIA (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
EPIDIDYMITIS (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
MENOMETRORRHAGIA (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
SCROTAL SWELLING (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 0 | 2 | 0
WOUND (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
LIMB INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 4 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
MUSCLE RUPTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
DEVICE BREAKAGE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
FRACTURED SACRUM (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
BURNS SECOND DEGREE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
PUBIC RAMI FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
DISLOCATION OF VERTEBRA (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
ABDOMINAL WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
MEDICAL DEVICE COMPLICATION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
DISLOCATION OF JOINT PROSTHESIS (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6 | 0
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
TENOSYNOVITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
LIMB DEFORMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 7 | 0
TENDON DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
FINGER DEFORMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
JOINT DESTRUCTION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
RHEUMATOID NODULE (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 18 | 2
OSTEOPOROTIC FRACTURE (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
MUSCULOSKELETAL DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 0
THROAT TIGHTNESS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
DEATH (General disorders) | 0 | 1 | 0 | 0
HERNIA (General disorders) | 1 | 0 | 1 | 0
PYREXIA (General disorders) | 0 | 0 | 1 | 0
CHEST PAIN (General disorders) | 1 | 4 | 2 | 0
SUDDEN DEATH (General disorders) | 0 | 0 | 1 | 0
CHEST DISCOMFORT (General disorders) | 0 | 0 | 1 | 0
IMPAIRED HEALING (General disorders) | 0 | 0 | 1 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 0 | 1 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | 0
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
OVARIAN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
BOWEN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
NEOPLASM PROSTATE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
LIGHT CHAIN DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 5 | 0
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 4 | 0
BENIGN SALIVARY GLAND NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
SMALL CELL LUNG CANCER STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aba 10mg/kg+MTX (N=115) | Aba 2mg/kg+MTX (N=105) | Abatacept (LT) (N=219) | Placebo+MTX (N=119)
CATARACT (Eye disorders) | 1 | 1 | 19 | 3
CONJUNCTIVITIS (Eye disorders) | 3 | 2 | 18 | 2
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 4 | 13 | 4
HYPERTENSION (Vascular disorders) | 8 | 12 | 45 | 9
ANXIETY (Psychiatric disorders) | 3 | 1 | 23 | 3
INSOMNIA (Psychiatric disorders) | 5 | 3 | 17 | 4
DEPRESSION (Psychiatric disorders) | 3 | 3 | 30 | 9
HEADACHE (Nervous system disorders) | 16 | 17 | 43 | 19
SCIATICA (Nervous system disorders) | 1 | 0 | 20 | 0
DIZZINESS (Nervous system disorders) | 6 | 5 | 32 | 3
PARAESTHESIA (Nervous system disorders) | 2 | 1 | 15 | 4
HYPOAESTHESIA (Nervous system disorders) | 2 | 4 | 13 | 1
NAUSEA (Gastrointestinal disorders) | 16 | 12 | 28 | 17
VOMITING (Gastrointestinal disorders) | 4 | 4 | 18 | 9
DIARRHOEA (Gastrointestinal disorders) | 14 | 11 | 40 | 9
DYSPEPSIA (Gastrointestinal disorders) | 7 | 12 | 31 | 7
CONSTIPATION (Gastrointestinal disorders) | 4 | 5 | 20 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 7 | 7 | 16 | 5
MOUTH ULCERATION (Gastrointestinal disorders) | 1 | 1 | 7 | 7
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 3 | 0 | 17 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 | 3 | 21 | 3
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 1 | 11 | 3
VERTIGO (Ear and labyrinth disorders) | 2 | 1 | 14 | 2
RHINITIS (Infections and infestations) | 2 | 1 | 19 | 0
INFLUENZA (Infections and infestations) | 5 | 3 | 23 | 6
SINUSITIS (Infections and infestations) | 5 | 7 | 50 | 10
BRONCHITIS (Infections and infestations) | 9 | 7 | 51 | 5
PHARYNGITIS (Infections and infestations) | 3 | 2 | 20 | 3
HERPES ZOSTER (Infections and infestations) | 3 | 2 | 25 | 0
TOOTH ABSCESS (Infections and infestations) | 2 | 2 | 11 | 3
GASTROENTERITIS (Infections and infestations) | 3 | 2 | 26 | 2
NASOPHARYNGITIS (Infections and infestations) | 17 | 19 | 76 | 11
FUNGAL INFECTION (Infections and infestations) | 2 | 3 | 12 | 3
LOCALISED INFECTION (Infections and infestations) | 0 | 1 | 11 | 1
URINARY TRACT INFECTION (Infections and infestations) | 3 | 2 | 48 | 3
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 1 | 18 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 13 | 10 | 58 | 9
HAEMATURIA (Renal and urinary disorders) | 0 | 1 | 13 | 0
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 13 | 0
RASH (Skin and subcutaneous tissue disorders) | 6 | 4 | 31 | 6
ECZEMA (Skin and subcutaneous tissue disorders) | 1 | 1 | 13 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 0 | 12 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 3 | 1 | 11 | 2
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 | 1 | 11 | 3
FALL (Injury, poisoning and procedural complications) | 2 | 0 | 16 | 2
CONTUSION (Injury, poisoning and procedural complications) | 2 | 2 | 15 | 1
BURSITIS (Musculoskeletal and connective tissue disorders) | 3 | 2 | 17 | 1
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 4 | 3 | 8 | 7
BACK PAIN (Musculoskeletal and connective tissue disorders) | 10 | 9 | 65 | 9
NECK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 2 | 21 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 | 10 | 30 | 11
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 | 3 | 16 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 2 | 11 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 3 | 19 | 4
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 6 | 15 | 4
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 35 | 50 | 100 | 55
COUGH (Respiratory, thoracic and mediastinal disorders) | 16 | 10 | 52 | 15
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 17 | 7
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 13 | 2
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 28 | 9
FATIGUE (General disorders) | 7 | 9 | 26 | 15
PYREXIA (General disorders) | 3 | 1 | 13 | 1
CHEST PAIN (General disorders) | 2 | 3 | 14 | 1
OEDEMA PERIPHERAL (General disorders) | 4 | 3 | 29 | 5
INFLUENZA LIKE ILLNESS (General disorders) | 1 | 2 | 12 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.